## Protocol I4V-MC-JAHL(a)

Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Baricitinib in Adult Patients with Moderate to Severe Atopic Dermatitis

NCT03334396

Approval Date: 15-Dec-2017

# Protocol I4V-MC-JAHL(a) A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Baricitinib in Adult Patients with Moderate to Severe Atopic Dermatitis

## **BREEZE-AD1**

EudraCT Number: 2017-000870-12

## **Confidential Information**

The information contained in this document is confidential and is intended for the use of clinical investigators. It is the property of Eli Lilly and Company or its subsidiaries and should not be copied by or distributed to persons not involved in the clinical investigation of baricitinib (LY3009104), unless such persons are bound by a confidentiality agreement with Eli Lilly and Company or its subsidiaries.

Note to Regulatory Authorities: This document may contain protected personal data and/or commercially confidential information exempt from public disclosure. Eli Lilly and Company requests consultation regarding release/redaction prior to any public release. In the United States, this document is subject to Freedom of Information Act (FOIA) Exemption 4 and may not be reproduced or otherwise disseminated without the written approval of Eli Lilly and Company or its subsidiaries.

## Baricitinib (LY3009104)

Study I4V-MC-JAHL is a Phase 3, multicenter, randomized, double-blind, placebo-controlled, parallel-group, outpatient, 25-week study designed to evaluate the efficacy and safety of baricitinib 1-mg, 2-mg, and 4-mg in patients with moderate to severe atopic dermatitis.

Eli Lilly and Company Indianapolis, Indiana USA 46285

Protocol Electronically Signed and Approved by Lilly: 29 Jun 2017 Amendment (a) Electronically Signed and Approved by Lilly on approval date provided below.

Approval Date: 15-Dec-2017 GMT

# **Table of Contents**

| Section | Page |
|---|---|
| 1. Synopsis | 9 |
| 2. Schedule of Activities | 13 |
| 3. Introduction | 18 |
| 3.1. Background | 18 |
| 3.2. Study Rationale | 19 |
| 3.3. Benefit/Risk Assessment | 19 |
| 4. Objectives and Endpoints | 20 |
| 5. Study Design | 22 |
| 5.1. Overall Design | |
| 5.1.1. Period 1: Screening | 22 |
| 5.1.2. Period 2: Double Blind Placebo-Controlled Treatment | 23 |
| 5.1.3. Period 3: Post-Treatment Follow-Up | 23 |
| 5.2. Number of Participants | 25 |
| 5.3. End of Study Definition | 25 |
| 5.4. Scientific Rationale for Study Design | |
| 5.5. Justification for Dose | |
| 5.5.1. Dose Adjustment for Renal Impairment | 26 |
| 6. Study Population | |
| 6.1. Inclusion Criteria | |
| 6.2. Exclusion Criteria | |
| 6.3. Lifestyle Restrictions | |
| 6.4. Screen Failures | |
| 7. Treatments | |
| 7.1. Treatments Administered | |
| 7.1.1. Packaging and Labeling | |
| 7.1.2. Medical Devices. | |
| 7.2. Method of Treatment Assignment | |
| 7.2.1. Selection and Timing of Doses. | |
| 7.2.2. Dose Adjustment for Renal Impairment | |
| 7.3. Blinding | |
| <ul><li>7.4. Dosage Modification</li><li>7.5. Preparation/Handling/Storage/Accountability</li></ul> | |
| 7.6. Treatment Compliance | |
| 7.7. Concomitant Therapy | |
| 7.7. Componition in the p J | |

| 7.7.1. P | rohibited Medications and Procedures | 39 |
|--------------|-------------------------------------------------------|-----|
| 7.7.2. P | ermitted Medications and Procedures | 40 |
| 7.7.3. R | escue Therapy | 41 |
| 7.8. Treatn | nent after the End of the Study | 42 |
| 7.8.1. S | tudy Extensions | 42 |
| 7.8.2. C | ontinued Access | 43 |
| 8. Discontin | uation Criteria | 44 |
| | ntinuation from Study Treatment | |
| | emporary Interruption from Investigational Product | |
| | ermanent Discontinuation from Investigational Product | |
| 8.1.3. D | Discontinuation of Inadvertently Enrolled Patients | 47 |
| | tinuation from the Study | |
| | Follow-Up | |
| 9. Study Ass | sessments and Procedures | 49 |
| | ey Assessments | |
| | rimary Efficacy Assessments | |
| | econdary Efficacy Assessments | |
| 9.1.2.1. | Eczema Area and Severity Index Scores | |
| 9.1.2.2. | SCORing Atopic Dermatitis | |
| 9.1.2.3. | Hospital Anxiety Depression Scale | |
| 9.1.3. H | lealth Outcomes and Quality-of-Life Measures | 50 |
| 9.1.3.1. | Patient-Oriented Eczema Measure | 50 |
| 9.1.3.2. | Itch Numeric Rating Scale | 50 |
| 9.1.3.3. | Nocturnal Sleep-Wake and Itch Patterns | 50 |
| 9.1.3.4. | Atopic Dermatitis Sleep Scale | 50 |
| 9.1.3.5. | Skin Pain Numeric Rating Scale | 50 |
| 9.1.3.6. | Patient Global Impression of Severity | 51 |
| 9.1.3.7. | Dermatology Life Quality Index | 51 |
| 9.1.3.8. | European Quality of Life–5 Dimensions–5 Levels | 51 |
| 9.1.3.9. | Work Productivity and Activity Impairment | |
| | Questionnaire—Atopic Dermatitis | |
| | ppropriateness of Assessments | |
| | se Events | |
| | erious Adverse Events. | |
| 9.2.1.1. | Suspected Unexpected Serious Adverse Reactions | |
| | dverse Events of Special Interest | |
| | omplaint Handling | |
| 44 Treatn | nent at Liverdage | 5.4 |

| 9.4. Safe | ety | 54 |
|-------------|-------------------------------------------------|----|
| 9.4.1. | Electrocardiograms | 54 |
| 9.4.2. | Vital Signs | 54 |
| 9.4.3. | Physical Exam | 55 |
| 9.4.4. | Laboratory Tests | 55 |
| 9.4.5. | Columbia Suicide Severity Rating Scale | 55 |
| 9.4.6. | Self-Harm and Follow-up Supplement Forms | 55 |
| 9.4.7. | Chest x-ray and Tuberculosis Testing. | 55 |
| 9.4.8. | Hepatitis B Virus DNA Monitoring | 56 |
| 9.4.9. | Hepatic Safety Monitoring and Data Collection | 56 |
| 9.4.10. | Safety Monitoring | 57 |
| 9.5. Pha | rmacokinetics | 57 |
| 9.6. Pha | rmacodynamics | 59 |
| 9.7. Pha | rmacogenetics | 59 |
| 9.7.1. | Blood Samples for Pharmacogenetic Research | 59 |
| 9.8. Bio | markers | 60 |
| 9.9. Med | dical Resource Utilization and Health Economics | 60 |
| 0. Statisti | cal Considerations | 61 |
| 10.1. San | ple Size Determination | 61 |
| | ulations for Analyses | |
| - | istical Analyses | |
| 10.3.1. | General Statistical Considerations | |
| 10.3.2. | Treatment Group Comparability | 64 |
| 10.3.2. | | |
| 10.3.2. | • | |
| 10.3.2. | 3. Concomitant Therapy | 64 |
| 10.3.2. | 4. Treatment Compliance | |
| 10.3.3. | Efficacy Analyses | |
| 10.3.3. | | |
| 10.3.3. | | |
| 10.3.4. | Safety Analyses | |
| 10.3.5. | Pharmacokinetic/Pharmacodynamic Analyses | |
| 10.3.6. | Other Analyses | |
| 10.3.6. | • | |
| 10.3.6. | | |
| 10.3.7. | Interim Analyses | |
| 10.3.7. | • | |
| | 2. Adjudication Committee | |

# Page 5

| 11. | References | 68 |
|-----|------------|----|
| 12. | Appendices | 72 |

# List of Tables

| Table | | Page |
|---|---|---|
| Table JAHL.1. | I4V-MC-JAHL Schedule of Activities | 13 |
| Table JAHL.2. | Objectives and Endpoints. | 20 |
| Table JAHL.3. | Treatment Regimens | 36 |
| Table JAHL.4. | Criteria for Temporary Interruption of Investigational Product | 44 |

# **List of Figures**

| Figure | Page | |
|---|---|---|
| Figure JAHL.1. | Illustration of study design for Clinical Protocol I4V-MC-JAHL | 24 |

# **List of Appendices**

| Appendix | | Page |
|---|---|---|
| Appendix 1. | Abbreviations and Definitions. | 73 |
| Appendix 2. | Clinical Laboratory Tests | 77 |
| Appendix 3. | Study Governance Considerations | 79 |
| Appendix 4. | Hepatic Monitoring Tests For Treatment-Emergent Abnormality | 83 |
| Appendix 5. | Liver Function Testing and Hepatic Safety Monitoring | 84 |
| Appendix 6. | American Academy of Dermatology: Criteria for the Diagnosis and Assessment of Atopic Dermatitis | 85 |
| Appendix 7. | Classification of Potency for Topical Corticosteroids | 86 |
| Appendix 8. | Protocol Amendment I4V-MC-JAHL(a) Summary - A Multicenter,<br>Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to<br>Evaluate the Efficacy and Safety of Baricitinib in Adult Patients with<br>Moderate to Severe Atopic Dermatitis | 87 |

# 1. Synopsis

#### Title of Study:

A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Baricitinib in Adult Patients with Moderate to Severe Atopic Dermatitis

#### Rationale:

Atopic dermatitis (AD) is a pruritic, chronic or chronically relapsing, highly symptomatic inflammatory skin disease characterized by excessive T cell activation leading to significant skin infiltration by T cells and dendritic cells (Bieber 2010). Presentation is varied, but includes skin manifestations and pruritus, with associated sleep disturbances and subsequent skin infections. The course of disease includes relapses of varying duration and severity.

Baricitinib is an orally available, selective Janus kinase (JAK) inhibitor with potency and selectivity for JAK1 and JAK2 and less potency for JAK3 or tyrosine kinase 2 (TYK2) (Fridman et al. 2010). The pathogenesis of AD is thought to be modulated through thymic stromal lymphopoietin (TSLP), interleukin (IL)-13, IL-4, IL-5, IL-22, and IL-31, many of which activate receptors with downstream signaling through intracellular JAK1/JAK2/TYK2 (Nomura and Kabashima 2015). This activity profile suggests that baricitinib would inhibit cytokines involved in AD pathogenesis.

Clinical studies have established that baricitinib is effective in autoimmune/autoinflammatory diseases involving the joints, kidneys, and skin. Baricitinib was effective at reducing swollen and tender joints in patients with rheumatoid arthritis (Genovese et al. 2016; Dougados et al. 2017; Fleischmann et al. 2017; Taylor et al. 2017); was effective at reducing disease severity in patients with moderate to severe plaque psoriasis (Papp et al. 2016); was effective at reducing the urinary albumin-to-creatinine ratio in patients with diabetic kidney disease (Tuttle et al. 2015); and in a recently completed Phase 2 study (I4V-MC-JAHG) was effective at reducing disease severity in patients with moderate to severe AD. The mechanism of action, combined with demonstration of clinical benefit in inflammatory diseases involving joints, kidneys, and skin, provides the rationale for evaluating baricitinib in moderate to severe AD.

#### **Objectives/Endpoints:**

| Objectives | Endpoints |
|---|---|
| Primary | |
| To test the hypothesis that baricitinib 4-mg QD or | <ul> <li>Proportion of patients achieving IGA of 0 or 1 with</li> </ul> |
| baricitinib 2-mg QD is superior to placebo in the | a $\geq$ 2-point improvement at Week 16. |
| treatment of patients with moderate to severe AD. | |
| Key Secondary | |
| These are prespecified objectives that will be adjusted | for multiplicity |
| To test the hypothesis that baricitinib 1-mg QD is | <ul> <li>Proportion of patients achieving IGA of 0 or 1 with</li> </ul> |
| superior to placebo in the treatment of patients with | a $\geq$ 2-point improvement at Week 16. |
| moderate to severe AD. | |

| Objectives | Endpoints |
|---|---|
| To compare the efficacy of baricitinib 1-mg QD, 2-mg QD, or 4-mg QD to placebo in AD during the 16-week double-blind placebo-controlled treatment period as measured by improvement in signs and symptoms of AD. | <ul> <li>Proportion of patients achieving EASI75 at 16 weeks</li> <li>Proportion of patients achieving EASI90 at 16 weeks</li> <li>Percent change from baseline in EASI score at 16 weeks</li> <li>Proportion of patients achieving SCORAD75 at 16 weeks.</li> </ul> |
| To compare the efficacy of baricitinib 1-mg QD, 2-mg QD, or 4-mg QD to placebo in AD during the 16-week double-blind placebo-controlled treatment period as assessed by patient-reported outcome measures. | <ul> <li>Proportions of patients achieving a 4-point improvement in Itch NRS at 1 week, 2 weeks, 4 weeks, and 16 weeks</li> <li>Mean change from baseline in the score of Item 2 of the ADSS at 1 week and 16 weeks</li> <li>Mean change from baseline in Skin Pain NRS at 16 weeks.</li> </ul> |
| Other Secondary Objectives | |
| These are prespecified objectives that will not be adjust. To test the hypothesis that baricitinib 1-mg QD, 2-mg QD, or 4-mg QD is superior to placebo in the treatment of patients with moderate to severe AD. To compare the efficacy of baricitinib 1-mg QD, | <ul> <li>Proportion of patients achieving IGA of 0 or 1 with a ≥2-point improvement at Week 4.</li> <li>Proportion of patients achieving EASI50 at</li> </ul> |
| 2-mg QD, or 4-mg QD to placebo in AD during the 16-week double-blind placebo-controlled period as measured by improvement in signs and symptoms of AD. | <ul> <li>16 weeks</li> <li>Proportion of patients achieving IGA of 0 at 16 weeks</li> <li>Mean change from baseline in SCORAD at 16 weeks</li> <li>Proportion of patients achieving SCORAD90 at 16 weeks</li> <li>Mean change from baseline in body surface area affected at 16 weeks</li> <li>Proportion of patients developing skin infections requiring antibiotic treatment by Week 16.</li> </ul> |
| To compare the efficacy of baricitinib 1-mg QD, 2-mg QD, or 4-mg QD to placebo in AD during the 16-week double-blind placebo-controlled treatment period as assessed by patient-reported outcome/QoL measures. | <ul> <li>Percent change from baseline in Itch NRS at 1 week and 16 weeks</li> <li>Mean change from baseline in Itch NRS at 4 weeks and 16 weeks</li> <li>Mean change from baseline in the total score of the POEM at 16 weeks</li> <li>Mean change in PGI-S-AD scores at 16 weeks</li> <li>Mean change from baseline in the HADS at 16 weeks</li> <li>Mean change in DLQI scores at 16 weeks</li> <li>Mean change in WPAI scores at 16 weeks</li> <li>Mean change in EQ-5D-5L scores at 16 weeks.</li> </ul> |

Abbreviations: AD = atopic dermatitis; ADSS = Atopic Dermatitis Sleep Scale; DLQI = Dermatology Life Quality Index; EASI = Eczema Area and Severity Index; EQ-5D-5L = the European Quality of Life-5 Dimensions-5 Levels; HADS = Hospital Anxiety Depression Scale; IGA = Investigator's Global Assessment; NRS = numeric rating scale; QD = once daily; PGI-S-AD = Patient Global Impression of Severity-Atopic Dermatitis; POEM = Patient-Oriented Eczema Measure; QoL = quality of life; SCORAD = SCORing Atopic Dermatitis; WPAI = Work Productivity and Activity Impairment.

#### **Summary of Study Design:**

Study I4V-MC-JAHL (JAHL) is a Phase 3, multicenter, randomized, double-blind, placebo-controlled, parallel-group, outpatient study evaluating the efficacy and safety of baricitinib 4-mg once daily (QD), 2-mg QD, and 1-mg QD as compared to placebo in adult patients with moderate to severe AD. The study population will include patients aged 18 years or older who have moderate to severe AD and a history of inadequate response or intolerance to existing topical therapies.

The study duration will be up to 25 weeks over 3 study periods:

- Period 1: Screening Period lasting from 8 to 35 days prior to Week 0 (baseline, Visit 2).
- Period 2: Double-Blinded Treatment Period, lasting from Week 0 (baseline, Visit 2) through Week 16 (Visit 8) inclusive:
  - At completion of the double-blind treatment period, eligible patients will be provided the option to participate in the long-term extension study I4V-MC-JAHN (JAHN). Those not eligible or who chose not to participate will proceed to the post-treatment follow-up period.
- Period 3: Post-Treatment Follow-Up Period, spanning the period from the last treatment visit at Week 16
  (Visit 8) or Early Termination Visit (ETV) to approximately 4 weeks following the last dose of
  investigational product.

#### **Treatment Arms and Duration:**

Patients will be randomized at Week 0 to 1 of 4 treatment groups: placebo once daily (QD), baricitinib 1-mg QD, baricitinib 2-mg QD, or baricitinib 4-mg QD. The study duration will be up to 25 weeks (Screening Period: up to 5 weeks prior to randomization; Double-Blinded Treatment Period: 16 weeks; Follow-up Period: approximately 4 weeks after the last dose of investigational product).

#### **Number of Patients:**

This study will include approximately 600 patients with AD who will be randomized 2:1:1:1 to placebo QD or 1 of 3 dose groups of baricitinib (1-mg QD, 2-mg QD, or 4-mg QD) (240 patients in the placebo arm; 120 patients in each baricitinib treatment group).

#### **Statistical Analysis:**

Unless otherwise specified, the efficacy and health outcome analyses will be conducted on the intent-to-treat population and safety analyses will be conducted on those patients who receive at least 1 dose of investigational product.

Treatment comparisons of discrete efficacy variables will be made using a logistic regression analysis with treatment, baseline disease severity, and region in the model. The proportions and 95% confidence interval (CI) will

be reported. If a patient needs to use rescue medication, the data after rescue onward will be considered missing and missing data will be imputed using the nonresponder imputation (NRI) method. All patients who discontinue the study or study treatment at any time for any reason will be defined as nonresponders for the NRI analysis for categorical variables after discontinuation onward. Additional analyses will be done using all observed data whether rescue medication was used or not.

Treatment comparisons of continuous efficacy and health outcome variables will be made using mixed-effects model of repeated measures (MMRM) with treatment, region, baseline severity, visit, and treatment-by-visit interaction as fixed categorical effects and baseline score and baseline score-by-visit interaction as fixed continuous effects. An unstructured covariance matrix will be used to model the within-patient variance—covariance errors. Type III sums of squares for the least squares means (LSMs) will be used for the statistical comparison and contrasts will be set up within the model to compare treatment groups at specific time points of interest.

Fisher exact test will be used for all adverse events (AEs), baseline, discontinuation, and other categorical safety data. Continuous vital signs and laboratory values will be analyzed by an analysis of covariance (ANCOVA) with treatment and baseline values in the model.

# 2. Schedule of Activities

Table JAHL.1. I4V-MC-JAHL Schedule of Activities

| | Screening | | Double-Blind, Placebo-Controlled | | | | | | Post-treatment<br>Follow-Up |
|---|---|---|---|---|---|---|---|---|---|
| 77 77 1 | Period 1 | | | | | | | Period 3 | |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 801a |
| Weeks from Randomization | | 0 | 1 | 2 | 4 | 8 | 12 | 16 or ET | |
| Days from Randomization | | 0 | 7 | 14 | 28 | 56 | 84 | 112 | |
| Visit tolerance interval (days) | -8 to -35 | | ±2 | ±2 | ±2 | ±4 | ±4 | ±4 | 28 ± 4 after last<br>dose |
| Procedure | | | | | | | | | |
| Inclusion and exclusion review | X | X | | | | | | | |
| Informed consent | X | | | | | | | | |
| Clinical Assessments | | | | | | | | | |
| Demographics | X | | | | | | | | |
| Medical History | X | | | | | | | | |
| Substance Use (alcohol, tobacco use) | X | | | | | | | | |
| Previous and current AD treatments | X | | | | | | | | |
| Weight | X | X | | | X | X | X | X | X |
| Height | | X | | | | | | | |
| Vital signs (BP and Pulse) | X | X | X | X | X | X | X | X | X |
| Physical examination | X | | | | | | | | |
| Symptom-directed physical examb | | X | X | X | X | X | X | X | X |
| 12-lead ECG (single) | X | | | | | | | | |
| Chest x-ray <sup>c</sup> (posterior-anterior view) | X | | | | | | | | |
| TB test <sup>d</sup> | X | | | | | | | | |
| Read PPD if applicable (48–72 hours post PPD) | Xe | | | | | | | | |
| Pre-existing Conditions | X | | | | | | | | |
| Adverse Events | | X | X | X | X | X | X | X | X |
| Concomitant Medication | X | X | X | X | X | X | X | X | X |
| Actigraphy devices dispensed | X | X | X | X | | | | | |
| Actigraphy devices returnedf | | X | X | X | X | | | | |

| | Screening Period 1 | | Double-Blind, Placebo-Controlled | | | | | | Post-treatment<br>Follow-Up<br>Period 3 |
|---|---|---|---|---|---|---|---|---|---|
| Visit Number | | 2 | Period 2 2 3 4 5 6 7 8 | | | | | | 801a |
| Weeks from Randomization | 1 | | | | _ | | 12 | 16 or ET | 801" |
| | | 0 | 7 | 14 | 4 | 8 | | | |
| Days from Randomization | | 0 | / | 14 | 28 | 56 | 84 | 112 | |
| Visit tolerance interval (days) | -8 to -35 | | ±2 | ±2 | ±2 | ±4 | ±4 | ±4 | $28 \pm 4$ after last dose |
| ePRO (patient diary) dispensed | X | X | X | X | X | X | X | Xg | |
| ePRO (patient diary) returnedf | | X | X | X | X | X | X | X | Xg |
| Randomization | | X | | | | | | | |
| IWRS | X | X | X | X | X | X | X | X | X |
| IP dispensed | | X | X | X | X | X | X | | |
| IP returned and compliance assessed | | | X | X | X | X | X | X | |
| Dispense rescue TCSh | | | X | X | X | X | X | X | |
| Weigh (tube with cap) and record returned rescue TCSh | | | | Х | X | X | X | X | X |
| Scales | | | | | | | | | |
| IGA | X | X | X | X | X | X | X | X | X |
| EASI | X | X | X | X | X | X | X | X | X |
| SCORAD | X | X | X | X | X | X | X | X | X |
| Health Outcome Measures and Other<br>Questionnaires <sup>i</sup> | | | | | | | | | |
| POEM | X | X | X | X | X | X | X | X | X |
| DLQI | X | X | X | X | X | X | | X | X |
| HADS | X | X | | X | X | X | | X | |
| EQ-5D-5L | | X | X | X | X | X | X | X | X |
| WPAI-AD | | X | X | X | X | X | X | X | X |
| Itch NRS | X | X | X | X | X | X | X | X | X |
| Skin Pain NRS | X | X | X | X | X | X | X | X | X |
| ADSS | X | X | X | X | X | X | X | X | X |
| PGI-S-AD | X | X | X | X | X | X | X | X | X |
| C-SSRSi/Self-Harm Supplement Form | X | X | X | X | X | X | X | X | X |
| Self-Harm Follow-up Formk | X | X | X | X | X | X | X | X | X |

| | Screening | Double-Blind, Placebo-Controlled | | | | | Post-treatment<br>Follow-Up | | |
|---|---|---|---|---|---|---|---|---|---|
| | Period 1 | | | | Perio | d 2 | | | Period 3 |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 801a |
| Weeks from Randomization | | 0 | 1 | 2 | 4 | 8 | 12 | 16 or ET | |
| Days from Randomization | | 0 | 7 | 14 | 28 | 56 | 84 | 112 | |
| Visit tolerance interval (days) | -8 to -35 | | ±2 | ±2 | ±2 | ±4 | ±4 | ±4 | 28 ± 4 after last<br>dose |
| Laboratory Assessment | | | | | | | | | |
| Clinical Chemistryl | X | X | | | X | X | X | X | X |
| Hematology | X | X | | | X | X | X | X | X |
| Lipids (fasting) <sup>m</sup> | | X | | | | | X | Xn | X |
| Serum Pregnancyo | X | | | | | | | | |
| FSHP | X | | | | | | | | |
| TSH | X | | | | | | | | |
| HIV | X | | | | | | | | |
| HCV antibodyq | X | | | | | | | | |
| HBV testing | X | | | | | | | | |
| HBV DNAr | X | | | | | | | X | |
| Urinalysis | X | X | | | X | X | X | X | X |
| Urine Pregnancyo | | X | | X | X | X | X | X | X |
| Pharmacogenetics: blood | | X | | | | | | | |
| Serum immunoglobulins | | X | | | X | | | X | |
| Exploratory storage samples (serum and plasma) | | X | | | X | | | X | |
| RNA and biomarkers: blood | | X | | | X | | | X | |
| Baricitinib plasma concentration (PK sample)s | | X | | | X | X | X | X | |

Abbreviations: AD = atopic dermatitis; ADSS = Atopic Dermatitis Sleep Scale; BP = blood pressure; C-SSRS = Columbia Suicide Severity Rating Scale 11 categories suicidal ideation/suicidal behavior; DLQI = Dermatology Life Quality Index; EASI = Eczema Area and Severity Index; ECG = electrocardiogram; eGFR = estimated glomerular filtration rate; EQ-5D-5L = the European Quality of Life-5 Dimensions-5 Levels; ET = early termination; ePRO = electronic patient-reported outcomes (device); ETV = early termination visit; FSH = follicle-stimulating hormone; HADS = Hospital Anxiety Depression Scale; HBcAb = hepatitis B core antibody; HBsAb = hepatitis B surface antibody; HBV = hepatitis B virus; HIV = human immunodeficiency virus; IGA = Investigator's Global Assessment; IP = investigational product; IWRS = interactive web-response system; NRS = numeric rating scale; PGI-S-AD = Patient Global Impression of Severity-Atopic Dermatitis; PK = pharmacokinetic; POEM = Patient-Oriented Eczema Measure; PPD = purified protein derivative; RNA = ribonucleic acid; SCORAD = SCORing Atopic Dermatitis; TB = tuberculosis; TCS = topical corticosteroids; TSH =thyroid-stimulating hormone; WPAI-AD = Work Productivity and Activity Impairment-Atopic Dermatitis.

- Patients who have discontinued IP but remain in the study for more than 28 days without IP can combine their Visit 8/ET visit with their Visit 801 (follow up visit).
- b The symptom-directed physical examination may be repeated at the investigator's discretion any time a patient presents with physical complaints.
- c A posterior—anterior chest x-ray will be performed at screening unless one has been performed within the past 6 months and the x-ray and reports are available.
- d TB test(s) including PPD, QuantiFERON®-TB Gold, and T SPOT®. See Exclusion Criterion [38] for description of TB testing. In countries where the QuantiFERON-TB Gold test or T-SPOT is available, either test may be used instead of the PPD TB test. The QuantiFERON-TB Gold test may be performed locally or centrally; the T-SPOT must be performed locally. (Note: Exception: Patients with a history of active or latent TB who have documented evidence of appropriate treatment, have no history of re-exposure since their treatment was completed, and have a screening chest x-ray with no evidence of active TB may be enrolled if other entry criteria are met. Such patients would not be required to undergo the protocol-specific TB testing but must have a chest x-ray at screening.)
- e If PPD testing was chosen to test for TB, then the patient must return and PPD test read 48 to 72 hours after Visit 1 (post-PPD).
- f Actigraphy devices and ePRO devices will need to be collected from screen fail patients.
- g For patients not entering Study JAHN, their JAHL patient diary will continue to be dispensed at the final visit and returned at Visit 801.
- h Only required if patient met rescue criteria.
- i The following measures (POEM, DLQI, PGI-S-AD, Itch NRS, Skin Pain NRS, ADSS, EQ-5D-5L, WPAI-AD) should be completed prior to any clinical assessments being performed on days when study visits occur.
- j Suicidal ideation and behavior subscales excerpt Adapted for the assessment of 11 preferred ideation and behavior categories.
- k The Self-Harm Follow-up Form is only required if triggered by the Self-Harm Supplement Form.
- 1 Clinical chemistry will include the following value calculated by the central laboratory from serum creatinine: estimated glomerular filtration rate (eGFR, calculated using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] Creatinine 2009 equation).
- m Fasting lipid profile: Patients should not eat or drink anything except water for 12 hours prior to sample collection. If a patient attends these visits in a nonfasting state, this will not be considered a protocol violation.
- $_{\mbox{\scriptsize n}}$  Only required for patients completing an ETV prior to completion of Visit 7 (Week 12).
- o For all women of childbearing potential, a serum pregnancy test (central laboratory) will be performed at Visit 1. Urine pregnancy tests (local laboratory) will be performed at Visit 2 and at all subsequent study visits after Visit 3. If required per local regulations and/or institutional guidelines, pregnancy testing can occur at other times during the study treatment period.

- p For female patients ≥40 and <60 years of age who have had a cessation of menses for at least 12 months, an FSH test will be performed to confirm nonchildbearing potential (FSH ≥40 mIU/mL).
- q For patients who are positive for HCV antibody, a follow-up test for HCV RNA will be performed automatically. Patients who are positive for HCV antibody and negative for HCV RNA may be enrolled.
- r Patients who are positive for HBcAb and negative for HBV DNA may be enrolled. Any enrolled patient who is HBcAb positive, regardless of HBsAb status or level, must undergo HBV DNA testing per the schedule (see Section 9.4.8).
- s See Section 9.5 for details. At Visit 2 (Week 0) patients will take their investigational product in the clinic and PK samples will be drawn 15 minutes and 1 hour postdose. Other Visit 2 baseline laboratory samples should be taken before administration of investigational product. At Visit 5 (Week 4), patients should take their investigational product at home prior to visiting the clinic and samples will be collected 2 to 4 hours after the dose is taken at home. At Visit 6 (Week 8) and Visit 7 (Week 12), patients will be asked to **not** take their oral investigational product prior to visiting the clinic and a sample will be collected at any time predose on the day of the clinic visit. If the patient has taken his/her oral dose prior to the visit, the sample may be drawn anytime postdose, and the inability to collect a predose sample will not be considered a protocol violation. For Visit 8 (Week 16), patients should take their investigational product at home prior to visiting the clinic and samples will be collected 4 to 6 hours after the dose is taken at home. For the ETV, a sample may be drawn anytime if the last dose of investigational product was taken within the last 48 hours. For visits where PK samples will be collected, the actual date and exact 24-hour clock time of sample collection as well as the date and time of the 2 doses prior to the sample being drawn should be recorded. At Visit 5 (Week 4) and Visit 8 (Week 16), these 2 doses should be the dose given the morning of the day of sample collection and the dose given the previous day. At Visit 6 (Week 8) and Visit 7 (Week 12), the 2 previous doses should be the dose taken yesterday and the dose taken the day before that. This sampling schedule should be followed as closely as possible; however, failure to take PK samples at these specified times will not be considered a protocol violation.

## 3. Introduction

## 3.1. Background

Atopic dermatitis (AD), also known as eczema or atopic eczema, is a common, chronic, relapsing, highly symptomatic inflammatory skin disease (Bieber 2010). Patients with AD may present with skin lesions that can be acute with oozing, crusted, eroded vesicles or papules on erythematous plaques. Patients may also present with lesions that have a subacute appearance, with thick and excoriated plaques, or chronic appearance, with lichenified, slightly pigmented, excoriated plaques (Bieber 2010). Atopic dermatitis causes pruritus attacks throughout the day, which is the primary source of morbidity in this disorder (Simpson 2012). Pruritus often leads to an "itch–scratch" cycle, further compromising the epidermal barrier and resulting in dry skin, microbial colonization, and secondary infections (Krakowski et al. 2008), with 36% of patients reporting that they often or always scratch until their skin bleeds (Langenbruch et al. 2014). Pruritus from AD can worsen at night, resulting in sleep disturbances, with approximately 27% of adult patients with AD experiencing sleep disturbance as a result of itching (Langenbruch et al. 2014). In adult patients with moderate to severe AD, sleep quality and latency were significantly associated with poor quality of life (QoL) (Yano et al. 2013).

In clinical practice, AD is classified as mild, moderate, or severe based on a variety of clinical features, including severity of skin lesions and pruritus, and extent of disease (body surface area [BSA] involved).

Until recently, there were no Food and Drug Administration (FDA)-approved systemic treatments for patients with moderate to severe AD, with the exception of systemic corticosteroids. In March 2017, Dupixent (dupilumab) injection, an IgG4 monoclonal antibody that inhibits interleukin (IL)-4 and IL-13, was approved by the FDA for this patient population. In the European Union, only cyclosporine has been approved for the treatment of patients with severe AD (Bieber and Straeter 2015). A recently completed Phase 2 study (I4V-MC-JAHG [JAHG]) evaluated the safety and efficacy of baricitinib (a Janus kinase [JAK] inhibitor) in AD and results showed significant improvement in disease severity compared to placebo and no new safety concerns were identified.

In addition to AD, baricitinib has also been studied in Phase 3 in patients with rheumatoid arthritis (RA) and in Phase 2 in patients with diabetic nephropathy, moderate to severe psoriasis, and systemic lupus erythematosus.

Through 04 June 2016, baricitinib has been studied in more than 450 healthy volunteers and 4200 patients have received baricitinib in clinical studies. Of these, more than 2400 patients have been treated with baricitinib for more than a year and more than 900 patients have been treated with baricitinib for more than 2 years at doses of 2-mg QD and/or 4-mg QD across the RA clinical program. Baricitinib has been administered as single doses ranging from 1- to 40-mg and as repeat oral doses ranging from 2- to 20-mg to healthy subjects. Baricitinib has also been administered to patients with RA at doses up to 15-mg daily for 4 weeks, 10-mg daily for 24 weeks, 8-mg daily for 76 weeks, and lower doses up to 4-mg daily for up to approximately 5 years.

## 3.2. Study Rationale

The underlying cause of AD is not completely understood. Loss of function mutations in the gene for *filaggrin* (filament aggregating protein), a key protein in terminal differentiation of the epidermis contributing to barrier function, has been identified as the strongest genetic risk factor for AD in European populations (Palmer et al. 2006). At a cellular level, AD is characterized by excessive T cell activation caused by genetic and environmental factors, leading to significant skin infiltration by T cells and dendritic cells. The cytokine thymic stromal lymphopoietin (TSLP) is thought to act as a master switch that triggers the initiation and maintenance of AD (Moniaga et al. 2013; Ziegler et al. 2013). Overexpression of TSLP in keratinocytes, the most prevalent cell type in the skin, triggers robust itch-evoked scratching and the development of an AD-like skin phenotype in mice (Li et al. 2005). In addition to directly inducing itch by activating sensory neurons in the skin, TSLP also enhances maturation and differentiation of dendritic cells and naive CD4+ T cells and induces production of Th2-related cytokines involved in AD pathogenesis (Wilson et al. 2013; Divekar and Kita 2015). Thymic stromal lymphopoietin and other key cytokines involved in AD pathogenesis, such as IL-13, IL-5, IL-22, and IL-31, signal through receptors associated with intracellular JAK1/JAK2/tyrosine kinase 2 (TYK2) signaling (Ziegler et al. 2013; Nomura and Kabashima 2015).

Janus kinases are a family of tyrosine kinases that mediate cytokine receptor signalling through phosphorylation and activation of signal transducers and activators of transcription (STAT) proteins. There are 4 known JAK family members: JAK1, JAK2, JAK3, and TYK2 (Clark et al. 2014). The relative affinity of JAK inhibitors for different members of the JAK kinase family allows for differentiation of JAK inhibitors in relation to their enzymatic inhibitory profile. In vitro assays indicate that baricitinib is a selective inhibitor of JAKs with potency and selectivity for JAK1/2 and less potency for JAK3 or TYK2 (Fridman et al. 2010). The balanced JAK1/JAK2 inhibitory profile of baricitinib suggests that baricitinib will have the greatest modulatory effect in cytokines signalling through a JAK1/JAK2 heterodimer intracellularly (or a JAK1/JAK2/TYK2), such as IL-6, TSLP, IL-13, or IL-31 (Vaddi and Luchi 2012).

The recently completed Phase 2 study of baricitinib in AD, JAHG, met its primary objective of proportion of patients achieving a 50% improvement from baseline in EASI scores compared to placebo. Baricitinib also showed statistically significant improvements for other disease severity analyses as well as multiple different patient-reported outcome (PRO) scales compared to placebo, further validating the hypothesis that JAK1/JAK2 signaling plays a key role in AD pathogenesis.

#### 3.3. Benefit/Risk Assessment

More information about the known and expected benefits, risks, serious adverse events (SAEs) and reasonably anticipated adverse events (AEs) of baricitinib are to be found in the Investigator's Brochure (IB).

# 4. Objectives and Endpoints

Table JAHL.2 shows the objectives and endpoints of the study.

Table JAHL.2. Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| To test the hypothesis that baricitinib 4-mg QD or baricitinib 2-mg QD is superior to placebo in the treatment of patients with moderate to severe AD. | • Proportion of patients achieving IGA of 0 or 1 with a ≥2-point improvement at Week 16. |
| Key Secondary These are prespecified objectives that will be adjusted | d for multiplicity |
| To test the hypothesis that baricitinib 1-mg QD is superior to placebo in the treatment of patients with moderate to severe AD. | <ul> <li>Proportion of patients achieving IGA of 0 or 1 with<br/>a ≥2-point improvement at Week 16.</li> </ul> |
| To compare the efficacy of baricitinib 1-mg QD, 2-mg QD, or 4-mg QD to placebo in AD during the 16-week double-blind placebo-controlled treatment period as measured by improvement in signs and symptoms of AD. | <ul> <li>Proportion of patients achieving EASI75 at 16 weeks</li> <li>Proportion of patients achieving EASI90 at 16 weeks</li> <li>Percent change from baseline in EASI score at 16 weeks</li> <li>Proportion of patients achieving SCORAD75 at 16 weeks.</li> </ul> |
| To compare the efficacy of baricitinib 1-mg QD, 2-mg QD, or 4-mg QD to placebo in AD during the 16-week double-blind placebo-controlled treatment period as assessed by patient-reported outcome measures. | <ul> <li>Proportions of patients achieving a 4-point improvement in Itch NRS at 1 week, 2 weeks, 4 weeks, and 16 weeks</li> <li>Mean change from baseline in the score of Item 2 of the ADSS at 1 week and 16 weeks.</li> <li>Mean change from baseline in Skin Pain NRS at 16 weeks.</li> </ul> |
| Other Secondary Objectives These are prespecified objectives that will not be adju | usted for multiplicity. |
| To test the hypothesis that baricitinib 1-mg QD, 2-mg QD, or 4-mg QD is superior to placebo in the treatment of patients with moderate to severe AD. | <ul> <li>Proportion of patients achieving IGA of 0 or 1 with<br/>a ≥2-point improvement at Week 4</li> </ul> |
| To compare the efficacy of baricitinib 1-mg QD, 2-mg QD, or 4-mg QD to placebo in AD during the 16-week double-blind placebo-controlled period as measured by physician-assessed signs and symptoms of AD. | <ul> <li>Proportion of patients achieving EASI50 at 16 weeks</li> <li>Proportion of patients achieving IGA of 0 at 16 weeks</li> <li>Mean change from baseline in SCORAD at 16 weeks</li> <li>Proportion of patients achieving SCORAD90 at 16 weeks</li> <li>Mean change from baseline in BSA affected at 16 weeks</li> <li>Proportion of patients developing skin infections requiring antibiotic treatment by Week 16.</li> </ul> |

| Objectives | Endpoints |
|---|---|
| To compare the efficacy of baricitinib 1-mg QD, 2-mg QD, or 4-mg QD to placebo in AD during the 16-week, double-blind, placebo-controlled treatment period as assessed by patient-reported outcome/QoL measures. | <ul> <li>Percent change from baseline in Itch NRS at 1 week and 16 weeks</li> <li>Mean change from baseline in Itch NRS at 4 weeks and 16 weeks</li> <li>Mean change from baseline in the total score of the POEM at 16 weeks</li> <li>Mean change in PGI-S-AD scores at 16 weeks</li> <li>Mean change from baseline in the HADS at 16 weeks</li> <li>Mean change in DLQI scores at 16 weeks</li> <li>Mean change in WPAI scores at 16 weeks</li> <li>Mean change in EQ-5D-5L scores at 16 weeks.</li> </ul> |

#### **Exploratory Objectives/Endpoints**

- Mean change from baseline in nocturnal itch assessed by actigraphy device at 1 week and 4 weeks
- Frequency of patient-reported "no itch" (Itch NRS score = 0) days from daily diaries from Week 12 to Week 16
- Frequency of patient-reported "no pain" (Skin Pain NRS score = 0) days from daily diaries from Week 12 to Week 16
- Mean change from baseline in the score of Item 1 of the ADSS at 1 week and 16 weeks
- Mean change from baseline in the score of Item 3 of the ADSS at 1 week and 16 weeks
- To evaluate changes from baseline in IgE levels during the study
- To evaluate changes from baseline in eosinophil levels during the study
- To characterize baricitinib pharmacokinetics in the AD population and explore relationships between baricitinib exposure and study endpoints.

Abbreviations: AD = atopic dermatitis; ADSS = Atopic Dermatitis Sleep Scale; BSA = body surface area; DLQI = Dermatology Life Quality Index; EASI = Eczema Area and Severity Index; EQ-5D-5L = the European Quality of Life-5 Dimensions-5 Levels; HADS = Hospital Anxiety Depression Scale; IgE = immunoglobulin E; IGA = Investigator's Global Assessment; NRS = numeric rating scale; QD = once daily; QoL = quality of life; PGI-S-AD = Patient Global Impression of Severity-Atopic Dermatitis; POEM = Patient-Oriented Eczema Measure; SCORAD = SCORing Atopic Dermatitis; WPAI = Work Productivity and Activity Impairment.

# 5. Study Design

## 5.1. Overall Design

Study I4V-MC-JAHL (JAHL) is a Phase 3, multicenter, randomized, double-blind, placebo-controlled, parallel-group, outpatient study evaluating the efficacy and safety of baricitinib 1-mg once daily (QD), 2-mg QD, and 4-mg QD as compared to placebo in adult patients with moderate to severe AD. The study is divided into 3 periods, a 5-week Screening period, a 16-week Double-Blinded Treatment period, and a 4-week Post-Treatment Follow-Up period. For those patients who complete the 16-week treatment period, there is an option to participate in the long-term extension study I4V-MC-JAHN (JAHN).

Approximately 600 patients ≥18 years of age who have responded inadequately to or who are intolerant to topical therapy will be randomized at a 2:1:1:1 ratio to receive placebo QD, baricitinib 1-mg QD, baricitinib 2-mg QD, or baricitinib 4-mg QD (240 patients in the placebo group; 120 patients in each baricitinib treatment group). Patients will be stratified at randomization according to disease severity (Investigator's Global Assessment [IGA] 3 vs. 4) and geographic region.

All procedures to be conducted during the study, including timing of all procedures, are indicated in the Schedule of Activities (Section 2). Section 9.4.4 describes collection of laboratory samples; Appendix 2, Appendix 4, and Appendix 5 list the specific laboratory tests that will be performed for this study. Study governance considerations are described in detail in Appendix 3. Section 10.3.7.1 outlines information regarding the data monitoring committee (DMC) and interim analyses.

# 5.1.1. Period 1: Screening

The duration of the Screening Period is between 8 and 35 days prior to Visit 2 (Week 0). At Visit 1, the patient will sign the informed consent form (ICF) prior to any study assessments, examinations, or procedures being performed (see Appendix 3). All screening procedures will be performed according to the Schedule of Activities (Section 2). Patients who receive a purified protein derivative (PPD) skin test at Visit 1 will need to return within 48 to 72 hours later to read the skin test. Prior to randomization, treatments for AD will be washed out: 4 weeks for systemic treatments and 2 weeks for topical treatments (not including emollients). Patients will be required to use emollients daily during the 14 days preceding randomization and throughout the study. If patients have been using emollients daily at the time of screening, then those cumulative days can be utilized to meet inclusion criterion [8]. Additionally, collection of data through daily diaries and actigraphy devices will be required throughout the screening period. The baseline for the daily PRO and actigraphy assessments will be the average score of the 7 days prior to randomization; thus, the minimum screening window was set at 8 days.

All patients who have not previously received the herpes zoster vaccine by screening will be encouraged (per local guidelines) to do so prior to randomization. Refer to the exclusion criterion [27] in Section 6 for additional information regarding herpes zoster vaccinations.

Patients who meet all of the inclusion and none of the exclusion criteria (Section 6) will continue to Visit 2

#### 5.1.2. Period 2: Double Blind Placebo-Controlled Treatment

At Visit 2 (Week 0, baseline), study eligibility for each patient will be reviewed, based on all inclusion and exclusion criteria (Section 6), and laboratory test results. Patients who meet all criteria will proceed to randomization and begin the 16-week double-blind, placebo-controlled treatment period.

At Visit 2, after laboratory samples are collected and all assessments are completed, patients will take the first dose of investigational product at the clinic and pharmacokinetic (PK) samples will be drawn 15 minutes and 1 hour postdose. Pharmacokinetic sampling and the related timing of dosing for investigational product for each visit are detailed in Section 9.5.

Patient will be randomized at a 2:1:1:1 ratio into 1 of the 4 treatment groups (placebo QD, baricitinib 1–mg QD, baricitinib 2–mg QD, or baricitinib 4–mg QD). Investigational product will be administered daily for 16 weeks (treatment period Visits 2 through 8; see Section 7). All patients will be required to use emollients daily. Daily diaries will continue to be utilized throughout the treatment period and through Week 4 for actigraphy devices. Download of this data will be required at study visits. The use of topical corticosteroids (TCS), topical calcineurin inhibitors (TCNIs), crisaborole, and systemic therapies for the treatment of AD are not allowed, except as part of rescue therapy for patients not responding to treatment. Details of rescue therapy and criteria are included in Section 7.7.3. Assessments of disease severity will be performed by the investigator at all study visits including unscheduled and early termination visits (ETVs).

The primary efficacy endpoint and final visit in the treatment period will be at Week 16 (Visit 8). Patients who complete through the Week 16 study visit will be eligible for inclusion in the long-term extension study JAHN (up to 2 additional years of treatment).

If a patient discontinues investigational product for any reason, the patient should remain in the study through Week 16 (Visit 8). If the patient refuses and wishes to withdraw consent, an ETV should be performed as soon as logistically possible.

# 5.1.3. Period 3: Post-Treatment Follow-Up

Patients who complete the study through Visit 8 (Week 16) and do not enter the long-term extension study will have a post-treatment follow-up visit (Visit 801) approximately 28 days after the last dose of investigational product.

Patients who have received at least 1 dose of investigational product and discontinue early from the study must have an ETV, and return for the post-treatment safety follow-up visit (Visit 801) approximately 28 days after the last dose of investigational product.

Patients who have discontinued investigational product but remain in the study for more than 28 days without investigational product will have an ETV if they chose to discontinue early; however, a separate follow-up visit (V801) is not required.

Patients should not initiate new systemic AD treatment during this period. However, if patients or investigators must initiate treatment, patients should complete an unscheduled visit prior to the first dose of the new therapy.

Figure JAHL.1 illustrates the study design. The 4 dosing regimens are described in Section 7.1. The blinding procedure is described in Section 7.3.



Abbreviations: AD = atopic dermatitis; eGFR = estimated glomerular filtration rate; PPD = purified protein derivative; QD = once daily; V = visit; W = week.

- <sup>a</sup> Applicable to patients taking topical treatments (excluding emollients) or systemic treatments for AD at the time of screening.
- <sup>b</sup> For patients randomized to the 4-mg QD dose who have renal impairment (defined as eGFR <60 mL/min/1.73 m<sup>2</sup>), the baricitinib dose will be 2-mg QD.
- c Patients for whom PPD skin test for the evaluation of tuberculosis infection was performed at V1 must return and PPD test must be read 48-72 hours after Visit 1 (post-PPD).
- <sup>d</sup> Occurs approximately 28 days after the last dose of IP. Not required for those patients entering the long-term extension study JAHN.

Figure JAHL.1. Illustration of study design for Clinical Protocol I4V-MC-JAHL.

## 5.2. Number of Participants

Approximately 600 participants will be enrolled; approximately 840 patients will be screened to achieve this enrollment.

# 5.3. End of Study Definition

End of the study is the date of the last visit or last scheduled procedure shown in the Schedule of Activities (Section 2) for the last patient.

# 5.4. Scientific Rationale for Study Design

This study will enroll moderate to severe AD patients with a history of inadequate response or intolerance to existing topical therapies for whom a systemic treatment such as baricitinib may therefore be appropriate.

During the screening period (Period 1), a washout of systemic and topical treatments for AD was incorporated prior to randomization to minimize confounding effects due to background treatment. The double-blind, placebo-controlled treatment period (Period 2) is designed to minimize bias in the evaluation of the efficacy and safety of 3 baricitinib doses, relative to placebo, through 16 weeks of treatment.

In consideration of the disease severity, all patients in Study JAHL are eligible for rescue to TCS. Investigators are allowed to rescue patients who are experiencing unacceptable or worsening symptoms of AD. Once rescue medication is used, the patient will be determined to be a nonresponder (See Section 7.7.3).

Investigator's Global Assessments are commonly used in clinical trials, both for qualifying patients for enrollment and for evaluating treatment efficacy (Langley et al. 2015; Futamura et al. 2016). There is no single "gold standard" disease severity scale for AD; however, IGA scales provide clinically meaningful measures to patients and investigators that are easily described and that correspond to disease severity categories (e.g., moderate to severe). The scale that will be used in this trial, the validated Investigator's Global Assessment of Atopic Dermatitis (vIGA-AD, referred to throughout the protocol as IGA), has been developed internally and assesses AD severity using a 5-point scale.

A 2:1:1:1 randomization scheme of placebo, 1-mg baricitinib, 2-mg baricitinib, and 4-mg baricitinib was implemented because increased placebo enrollment across treatment groups has been reported to decrease placebo response and to also increase statistical power (Mallinckrodt 2011).

The 16-week efficacy endpoint was chosen because it is likely that a robust clinical effect will be observed with baricitinib within this timeframe based on the Phase 2 study results in AD and from previous studies in another inflammatory skin condition.

The Post-Treatment Follow-Up Period (Period 3) is for safety monitoring after the patient has been off investigational product for approximately 28 days.

#### 5.5. Justification for Dose

The doses proposed for AD Phase 3 studies are baricitinib 1-mg, 2-mg, and 4-mg QD. These doses were chosen primarily based on the recently completed Phase 2 AD study, JAHG, and are additionally supported by PK, safety, and efficacy data for baricitinib in Phase 2 and Phase 3 RA studies and a Phase 2 psoriasis study.

In the Phase 2 Study JAHG, both the 2-mg and 4-mg doses showed benefit on the primary and major secondary endpoints (EASI, IGA, SCORAD, POEM and DLQI) as compared to placebo, and both doses had an acceptable safety profile at Week 16. However, the 4-mg dose appeared to demonstrate a more rapid benefit (at 4 weeks) on the more stringent endpoints (EASI75, EASI90, and IGA 0 or 1) compared to 2-mg dose particularly in the subgroup of patients with baseline EASI scores ≥16. The 4-mg dose resulted in statistically significant improvement in these endpoints at Week 4 and this level of response was maintained through Week 16. A similar trend between the baricitinib 4-mg and 2-mg doses was observed in patients with RA. Although in Study JAHG the 4-mg dose seemed to perform better than the 2-mg dose on more stringent endpoints, on other endpoints, including EASI-50, and EASI change from baseline, 2-mg and 4-mg doses showed similar efficacy compared to placebo. Thus based on available data, 3 doses will be included in Phase 3, including a 1-mg dose, to cover the range of exposures where clinical responses could be anticipated

## 5.5.1. Dose Adjustment for Renal Impairment

Baricitinib exposure increases with decreased renal function. Based on PK simulations of baricitinib exposures for the mild and moderate categories of renal function (stratified as estimated glomerular filtration rate [eGFR] 60 to <90 mL/min/1.73 m² and eGFR 30 to <60 mL/min/1.73 m², respectively), dose adjustment is not required for patients with eGFR ≥60 mL/min/1.73 m². Patients with eGFR <60 mL/min/1.73 m² who are randomized to the 4-mg dose will receive a dose of 2-mg QD, which will ensure that exposures do not exceed those of the 4-mg QD dose in patients with eGFR ≥60 mL/min/1.73 m². For patients randomized to the 2-mg dose or 1-mg dose, there will be no dose adjustment based on renal function. The dose adjustment for renal impairment will be managed by interactive web-response system (IWRS) to ensure maintenance of the treatment blind. This study will not enroll patients with screening eGFR <40 mL/min/1.73 m². See Section 8.1.1 for eGFR thresholds that trigger interruption of investigational product.

The procedure of dose adjustment based on renal function (eGFR) during the study is detailed in Section 7.2.2.

# 6. Study Population

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, are not permitted.

Study investigator(s) will review patient history and screening test results at Visit 1 and Visit 2 to determine if the patient meets all inclusion and none of the exclusion criteria to qualify for randomization in the study. All screening activities must be completed and reviewed before the patient is randomized.

## 6.1. Inclusion Criteria

#### **Informed Consent**

- [1] are at least 18 years of age at the time of informed consent.
  - Note: Use local requirements to provide consent if the age of adulthood is defined as >18 years
- [2] are able to read, understand, and give documented (electronic or paper signature) informed consent.

## **Type of Patient and Disease Characteristics**

- [3] have a diagnosis of AD at least 12 months prior to screening, as defined by the American Academy of Dermatology: Guidelines of care for the management of AD; Section 1. Diagnosis and assessment of atopic dermatitis (see Appendix 6).
- [4] have moderate to severe AD, including all of the following:
  - a. Eczema Area and Severity Index (EASI) score ≥16 at screening (Visit 1) and at randomization (Visit 2)
  - b. IGA score of  $\geq 3$  at screening (Visit 1) and at randomization (Visit 2)
  - c. ≥10% of BSA involvement at screening (Visit 1) and at randomization (Visit 2).
- [5] have a documented history by a physician and/or investigator of inadequate response to existing topical medications within 6 months preceding screening, or history of intolerance to topical therapy as defined by at least 1 of the following:
  - a. inability to achieve good disease control defined as mild disease or better (e.g., IGA ≤2) after use of at least a medium potency TCS for at least 4 weeks, or for the maximum duration recommended by the product prescribing information (e.g., 14 days for super-potent TCS), whichever is shorter. Topical corticosteroids may be used with or without TCNIs.

- b. Patients who failed systemic therapies intended to treat AD within 6 months preceding screening, such as cyclosporine, methotrexate, azathioprine, and mycophenolate mofetil will also be considered as a surrogate for having inadequate response to topical therapy.
- c. documented history of clinically significant adverse reactions with the use of TCS such as skin atrophy, allergic reactions, systemic effects that in the opinion of the investigator outweigh the benefits of retreatment.
- [6] agree to discontinue use of the following excluded medications/treatments for at least 4 weeks prior to randomization (Visit 2) and throughout the study:
  - a. oral systemic corticosteroids and leukotriene inhibitors
  - b. systemic immunomodulators, including, but not limited to, cyclosporine, methotrexate, mycophenolate mofetil, and azathioprine
  - c. sedating antihistamines, including, but not limited to, alimemazine, chlorphenamine, clemastine, cyproheptadine, diphenhydramine, hydroxyzine, ketotifen, and promethazine
    - Note: Patients may use newer, less sedating antihistamines (e.g., fexofenadine, loratadine, cetirizine).
  - d. any other systemic therapy used to treat AD or symptoms of AD (approved or off-label use)
  - e. phototherapy, includes therapeutic phototherapy (psoralen plus ultraviolet-A, ultraviolet-B), excimer laser as well as self-treatment with tanning beds.
- [7] agree to discontinue use of the following excluded medications for at least 2 weeks prior to randomization (Visit 2) and throughout the study:
  - a. TCS or topical immune modulators (e.g., tacrolimus or pimecrolimus)
  - b. Topical phosphodiesterase type 4 (PDE-4) inhibitor (crisaborole)
- [8] have applied emollients daily for at least 14 days prior to randomization and agree to use emollient daily throughout the treatment period.
- [9] Patients who are receiving chronic treatments to improve sleep should be on a stable dose for at least 2 weeks prior to screening as determined by the investigator. Sedating antihistamines (see above) are not permitted.

#### **Patient Characteristics**

- [10] are male or nonpregnant, nonbreastfeeding female patients, except
  - a. Male patients must agree to use 2 forms of birth control (1 must be highly effective, see below) while engaging in sexual intercourse with female partners of childbearing potential while enrolled in the study and for at least 4 weeks following the last dose of investigational product.

b. Female patients of childbearing potential must agree to use 2 forms of birth control, when engaging in sexual intercourse with a male partner while enrolled in the study and for at least 4 weeks following the last dose of investigational product.

The following birth control methods are considered acceptable (the patient should choose 2 to be used with their male partner, and 1 must be highly effective):

- highly effective birth control methods: oral, injectable, or implanted hormonal contraceptives (combined estrogen/progesterone or progesterone only, associated with inhibition of ovulation); intrauterine device or intrauterine system (e.g., progestin-releasing coil); or vasectomized male (with appropriate post-vasectomy documentation of the absence of sperm in the ejaculate).
- effective birth control methods: condom with a spermicidal foam, gel, film, cream, or suppository; occlusive cap (diaphragm or cervical/vault caps) with a spermicidal foam, gel, film, cream, or suppository; or oral hormonal contraceptives.

Note: When local guidelines concerning highly effective or effective methods of birth control differ from the above, the local guidelines must be followed.

- c. Females of nonchildbearing potential are not required to use birth control and they are defined as:
  - o women ≥60 years of age or women who are congenitally sterile, or
  - o women ≥40 and <60 years of age who have had a cessation of menses for ≥12 months and a follicle-stimulating hormone (FSH) test confirming nonchildbearing potential (≥40 mIU/mL or ≥40 IU/L), or women who are surgically sterile (i.e., have had a hysterectomy or bilateral oophorectomy or tubal ligation).

## 6.2. Exclusion Criteria

Patients will be excluded from study enrollment if they meet any of the following criteria:

## **Medical Conditions Related to Atopic Dermatitis**

- [11] are currently experiencing or have a history of other concomitant skin conditions (e.g., psoriasis or lupus erythematosus) that would interfere with evaluations of the effect of study medication on AD.
- [12] patients who, in the opinion of the investigator, are currently experiencing or have a history of erythrodermic, refractory, or unstable skin disease that requires frequent hospitalizations and/or intravenous treatment for skin infections that may interfere with participation in the study.
- [13] a history of eczema herpeticum within 12 months prior to screening.
- [14] a history of 2 or more episodes of eczema herpeticum in the past.

- [15] patients who are currently experiencing a skin infection that requires treatment, or is currently being treated, with topical or systemic antibiotics.
  - Note: Patients may not be rescreened until at least 4 weeks after the date of their previous screen failure and at least 2 weeks after resolution of the infection.
- [16] have any serious concomitant illness that is anticipated to require the use of systemic corticosteroids or otherwise interfere with study participation or require active frequent monitoring (e.g., unstable chronic asthma).
- [17] have been treated with the following therapies:
  - a. monoclonal antibody (e.g., ustekinumab, omalizumab, dupilumab) for less than 5 half-lives prior to randomization.
  - b. received prior treatment with any oral JAK inhibitor (e.g., tofacitinib, ruxolitinib) less than 4 weeks prior to randomization
  - c. received any parenteral corticosteroid administered by intramuscular or intravenous injection within 2 weeks prior to study entry (Visit 1) or within 6 weeks prior to planned randomization (Visit 2) or are anticipated to require parenteral injection of corticosteroids during the study.
  - d. have had an intra-articular corticosteroid injection within 2 weeks prior to study entry (Visit 1) or within 6 weeks prior to planned randomization (Visit 2).

Note: Intranasal or inhaled steroid use is allowed during the trial.

e. probenecid at the time of randomization (Visit 2) that cannot be discontinued for the duration of the study

#### **Medical Conditions in General**

- [18] are largely or wholly incapacitated permitting little or no self-care, such as being bedridden.
- [19] have uncontrolled arterial hypertension characterized by a repeated systolic blood pressure >160 mm Hg or diastolic blood pressure >100 mm Hg in a seated position.
- [20] have had any major surgery within 8 weeks prior to screening or will require major surgery during the study that, in the opinion of the investigator in consultation with Lilly or its designee, would pose an unacceptable risk to the patient if participating in the trial.
- [21] are immunocompromised and, in the opinion of the investigator, at an unacceptable risk for participating in the study.

- [22] have experienced any of the following within 12 weeks of screening: venous thromboembolic event (VTE), myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage III/IV heart failure.
- [23] have a history of recurrent (≥2) VTE or are considered at high risk of VTE as deemed by the investigator.
- [24] have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute an unacceptable risk when taking investigational product or interfere with the interpretation of data.
- [25] have a history of lymphoproliferative disease; or have signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly; or have active primary or recurrent malignant disease; or have been in remission from clinically significant malignancy for less than 5 years.
  - a. Patients with cervical carcinoma in situ that has been appropriately treated with no evidence of recurrence or metastatic disease for at least 3 years may participate in the study.
  - b. Patients with basal cell or squamous epithelial skin cancers that have been appropriately treated with no evidence of recurrence for at least 3 years may participate in the study.
- [26] have a current or recent clinically serious viral, bacterial, fungal, or parasitic infection, including but not limited to the following:
  - Note: A recent viral upper respiratory tract infection or uncomplicated urinary tract infection should not be considered clinically serious.
  - a. symptomatic herpes zoster infection within 12 weeks prior to screening.
  - b. a history of disseminated/complicated herpes zoster (e.g., multidermatomal involvement, ophthalmic zoster, CNS involvement, or post-herpetic neuralgia).
  - c. symptomatic herpes simplex at the time of randomization.
  - d. active or chronic viral infection from hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
  - e. household contact with a person with active tuberculosis (TB) and did not receive appropriate and documented prophylaxis for TB.
  - f. evidence of active TB or have previously had evidence of active TB and did not receive appropriate and documented treatment.
  - g. clinically serious infection or received intravenous antibiotics for an infection, within the past 4 weeks of randomization.

- h. any other active or recent infection within 4 weeks of randomization that, in the opinion of the investigator, would pose an unacceptable risk to the patient if participating in the study.
- [27] have been exposed to a live vaccine within 12 weeks prior to planned randomization or are expected to need/receive a live vaccine during the course of the study (with the exception of herpes zoster vaccination).
  - Note: Patients eligible for herpes zoster vaccine, who have not received it prior to screening will be encouraged (per local guidelines) to do so prior to randomization; vaccination must occur >4 weeks prior to randomization and start of investigational product. Patients will be excluded if they were exposed to herpes zoster vaccination within 4 weeks of planned randomization. Investigators should review the vaccination status of their patients and follow the local guidelines for vaccination of those ≥18 years of age with nonlive vaccines intended to prevent infectious disease prior to entering patients into the study.
- [28] have a history of chronic alcohol abuse, IV drug abuse, or other illicit drug abuse within the 2 years prior to screening.
- [29] presence of significant uncontrolled neuropsychiatric disorder, are clinically judged by the investigator to be at risk for suicide, or have a "yes" answer to any of the following:
  - a. Question 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) on the "Suicidal Ideation" portion of the Columbia Suicide Severity Rating Scale (C-SSRS) or
  - b. Question 5 (Active Suicidal Ideation with Specific Plan and Intent) on the "Suicidal Ideation" portion of the C-SSRS or
  - c. Any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act or behavior) on the "Suicidal Behavior" portion of the C-SSRS;

and the ideation or behavior occurred within 2 months prior to Visit 1.

**Note:** a patient does not necessarily have to be excluded if they have self-injurious behavior that would be classified as nonsuicidal self-injurious behavior. If this situation arises, the subject should be referred to a psychiatrist or appropriately trained professional as indicated.

[30] have donated more than a single unit of blood within 4 weeks prior to screening or intend to donate blood during the course of the study.

#### **Other Exclusions**

[31] are unable or unwilling to make themselves available for the duration of the study and/or are unwilling to follow study restrictions/procedures.

- [32] are currently enrolled in any other clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
- [33] have participated within the last 30 days in a clinical study involving an investigational product. If the previous investigational product has a long half-life (2 weeks or longer), at least 3 months or 5 half-lives (whichever is longer) should have passed.
- [34] have previously been randomized in this study or any other study investigating baricitinib.
- [35] are investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
- [36] are Lilly or Incyte employees or their designee.

#### **Diagnostic Assessments**

- [37] have screening electrocardiogram (ECG) abnormalities that, in the opinion of the investigator, are clinically significant and indicate an unacceptable risk for the patient's participation in the study.
- [38] have evidence of active TB or latent TB
  - a. have evidence of active TB, defined in this study as the following:
    - o documented by a positive PPD test (≥5 mm induration between approximately 48 and 72 hours after application, regardless of vaccination history), medical history, clinical features, and abnormal chest x-ray at screening.
    - o The QuantiFERON®-TB Gold test or T-SPOT®.TB test (as available and if compliant with local TB guidelines) may be used instead of the PPD test. Patients are excluded from the study if the test is not negative and there is clinical evidence of active TB.

Exception: Patients with a history of active TB who have documented evidence of appropriate treatment, have no history of re-exposure since their treatment was completed, and have a screening chest x-ray with no evidence of active TB may be enrolled if other entry criteria are met. Such patients would not be required to undergo the protocol-specific TB testing for PPD, QuantiFERON®-TB Gold test, or T-SPOT® TB test but must have a chest x-ray at screening.

- b. have evidence of untreated/inadequately or inappropriately treated latent TB, defined in this study as the following:
  - o documented to have a positive PPD test (≥5 mm induration between approximately 48 and 72 hours after application, regardless of vaccination history), no clinical features consistent with active TB, and a chest x-ray with no evidence of active TB at screening; or

- o PPD test is positive and the patient has no medical history or chest x-ray findings consistent with active TB, the patient may have a QuantiFERON®-TB Gold test or T-SPOT® TB test (as available and if compliant with local TB guidelines). If the test results are not negative, the patient will be considered to have latent TB (for purposes of this study); or
- QuantiFERON®-TB Gold test or T-SPOT® TB test (as available and if compliant with local TB guidelines) may be used instead of the PPD test. If the test results are positive, the patient will be considered to have latent TB. If the test is not negative, the test may be repeated once within approximately 2 weeks of the initial value. If the repeat test results are again not negative, the patient will be considered to have latent TB (for purposes of this study).

Exception: Patients who have evidence of latent TB may be enrolled if he or she completes at least 4 weeks of appropriate treatment prior to randomization and agrees to complete the remainder of treatment while in the trial.

Exception: Patients with a history of latent TB who have documented evidence of appropriate treatment, have no history of re-exposure since their treatment was completed, and have a screening chest x-ray with no evidence of active TB may be enrolled if other entry criteria are met. Such patients would not be required to undergo the protocol-specific TB testing for PPD, QuantiFERON®-TB Gold test, or T-SPOT® TB test but must have a chest x-ray at screening.

- [39] have a positive test HBV infection defined as:
  - a. positive for hepatitis B surface antigen (HBsAg), or
  - b. positive for hepatitis B core antibody (HBcAb) and positive hepatitis B virus deoxyribonucleic acid (HBV DNA).

Note: Patients who are HBcAb positive and HBV DNA negative may be enrolled in the study. Patients who meet these criteria at screening will be identified by the central laboratory and monitored during the study.

- [40] have HCV infection (positive for anti-hepatitis C antibody with confirmed presence of HCV ribonucleic acid (RNA)
  - Note: Patients who have documented anti-HCV treatment for a past HCV infection AND are HCV RNA negative may be enrolled in the study.
- [41] have evidence of HIV infection and/or positive HIV antibodies.
- [42] have screening laboratory test values, including thyroid-stimulating hormone (TSH), outside the reference range for the population or investigative site that, in the opinion of the investigator, pose an unacceptable risk for the patient's participation in the study.

Note: Patients who are receiving thyroxine as replacement therapy may participate in the study, provided stable therapy has been administered for ≥12 weeks and TSH is within the laboratory's reference range. Patients who are receiving stable thyroxine replacement therapy who have TSH marginally outside the laboratory's normal reference range may participate if the treating physician has documented that the thyroxine replacement therapy is adequate for the patient.

- [43] have any of the following specific abnormalities on screening laboratory tests:
  - a. AST or ALT >2x ULN
  - b. alkaline phosphatase (ALP)  $\geq 2x$  ULN
  - c. total bilirubin ≥1.5x ULN
  - d. hemoglobin <10.0 g/dL (100.0 g/L)
  - e. total white blood cell count <2500 cells/ $\mu$ L (<2.50x10<sup>3</sup>/ $\mu$ L or <2.50 GI/L)
  - f. neutropenia (absolute neutrophil count [ANC] <1200 cells/ $\mu$ L) (<1.20x10<sup>3</sup>/ $\mu$ L or <1.20 GI/L)
  - g. lymphopenia (lymphocyte count <750 cells/ $\mu$ L) (<0.75x10<sup>3</sup>/ $\mu$ L or <0.75 GI/L)
  - h. thrombocytopenia (platelets  $<100,000/\mu$ L) ( $<100x10^3/\mu$ L or <100 GI/L)
  - i. eGFR <40 mL/min/1.73 m<sup>2</sup> (Chronic Kidney Disease Epidemiology Collaboration equation [CKD-EPI] Creatinine 2009 equation).

Note: For cases with any of the aforementioned laboratory abnormalities (Exclusion Criteria [42] and [43]), the tests may be repeated during screening, and values resulting from repeat testing may be accepted for enrollment eligibility if they meet the eligibility criterion.

# 6.3. Lifestyle Restrictions

Not applicable.

## 6.4. Screen Failures

Patients who are entered into the study but do not meet the eligibility criteria for participation in this study (screen failure) may be rescreened a maximum of 2 times. If patients are rescreened, rescreening cannot occur until at least 4 weeks after the date of their previous screen failure. When rescreening is performed, the individual must sign a new ICF and will be assigned a new identification number. Additionally, all necessary screening procedures must be conducted at rescreen to ensure all eligibility criteria are met.
## 7. Treatments

#### 7.1. Treatments Administered

This study involves a comparison of placebo, baricitinib 1-mg, baricitinib 2-mg, and baricitinib 4-mg administered orally once a day. Table JAHL.3 shows the treatment regimens.

Table JAHL.3. Treatment Regimens

| Regimen | Investigational Product Supplied | Dose |
|----------------------|----------------------------------|-------------------|
| Baricitinib 4-mg QDa | Baricitinib 4-mg tablets | 3 tablets per day |
| | Placebo to match 2-mg tablets | |
| | Placebo to match 1-mg tablets | |
| Baricitinib 2–mg QD | Baricitinib 2-mg tablets | 3 tablets per day |
| | Placebo to match 4-mg tablets | |
| | Placebo to match 1-mg tablets | |
| Baricitinib 1-mg QD | Baricitinib 1-mg tablets | 3 tablets per day |
| | Placebo to match 4-mg tablets | |
| | Placebo to match 2-mg tablets | |
| Placebo QD | Placebo to match 4-mg tablets | 3 tablets per day |
| | Placebo to match 2-mg tablets | |
| | Placebo to match 1-mg tablets | |

Abbreviation: QD =once daily.

The investigator or his or her designee is responsible for the following:

- explaining the correct use of the investigational agent(s) to the patient
- verifying that instructions are followed properly
- maintaining accurate records of investigational product dispensing and collection
- at the end of the study, returning all unused medication to Lilly, or its designee, unless the sponsor and sites have agreed all unused medication is to be destroyed by the site, as allowed by local law.

# 7.1.1. Packaging and Labeling

The sponsor (or its designee) will provide the following investigational products:

- tablets containing 4-mg of baricitinib
- tablets containing 2-mg of baricitinib
- tablets containing 1-mg of baricitinib
- placebo tablets to match baricitinib 4-mg tablets, 2-mg tablets, and 1-mg tablets.

Packaging for each dose will include 3 tablets per day. Each tablet has a distinctive shape and color, 4-mg vs. 2-mg vs. 1-mg, and each strength tablet has a matching placebo. Each active

<sup>&</sup>lt;sup>a</sup> The baricitinib dose for patients randomized to the 4-mg QD treatment group who have renal impairment (defined as eGFR <60 mL/min/1.73 m<sup>2</sup>) will be 2-mg QD.

dose package will contain the appropriate active strength tablet, and corresponding placebo tablets for the other strengths, as noted in Table JAHL.3.

Investigational product tablets will be provided in blister packs.

Clinical trial materials will be labeled according to the country's regulatory requirements.

#### 7.1.2. Medical Devices

An actigraphy device, a hypoallergenic device worn on the wrist, will be used to collect sleep/wake patterns and quantify nocturnal scratching events. Each patient will be dispensed 2 actigraphy devices. One should be worn on the wrist during waking hours and the other should be worn only during hours of sleep. Patients will be provided instructions on use and when to bring the devices back to study site based on Schedule of Activities (Section 2). If devices are not worn as instructed, it will not be considered a protocol violation.

## 7.2. Method of Treatment Assignment

Patients who meet all criteria for enrollment will be randomized in a 2:1:1:1 ratio (placebo, baricitinib 1-mg; baricitinib 2-mg; baricitinib 4-mg) to double-blind treatment at Visit 2 (Week 0). Randomization will be stratified by geographic region (Europe [EU], Japan [JPN], rest-of-world [ROW]) and disease severity at baseline (IGA 3 vs. 4). Assignment to treatment groups will be determined by a computer-generated random sequence using an IWRS. The IWRS will be used to assign blister packs, each containing double-blind investigational product tablets to each patient, starting at Visit 2 (Week 0), and at each visit up to and including Visit 7 (Week 12). Site personnel will confirm that they have located the correct blister packs by entering a confirmation number found on the blister packs into the IWRS.

# 7.2.1. Selection and Timing of Doses

The investigational product (3 tablets from blister pack) should be taken once daily without regard to food and, if possible, at approximately the same time every day, usually at the start of the patient's day, to aid patient compliance. Refer to Section 9.5, Pharmacokinetics, for specific instructions on dose timing at certain visits where a PK sample is drawn.

# 7.2.2. Dose Adjustment for Renal Impairment

The rationale of dose adjustment for patients with documented renal impairment (defined as screening eGFR  $\geq$ 40 to <60 mL/min/1.73 m<sup>2</sup>) is detailed in Section 5.5.1.

The dose adjustment for renal impairment will be managed by IWRS to ensure maintenance of the treatment blind. The eGFR value from the screening visit (Visit 1) will be entered into IWRS at Visit 2, and IWRS will assign the treatment doses accordingly.

Patients with documented renal impairment (defined as screening eGFR  $\geq$ 40 to <60 mL/min/1.73 m<sup>2</sup>), who are randomized to the 4-mg active treatment arm will receive a dose of 2-mg QD by the IWRS. For patients randomized to the 2-mg dose or 1-mg dose, there will be no dose adjustment based on renal function.

No dose adjustment will be made for patients with screening eGFR ≥60 mL/min/1.73 m<sup>2</sup>. These patients who are randomized to active treatment will receive their assigned dose, either baricitinib 4–mg, 2–mg, or 1–mg, respectively.

During the study, for patients with documented renal impairment when the subsequent eGFR falls <30 mL/min/1.73 m², investigational product will be withheld until their eGFR becomes ≥40 mL/min/1.73 m², whereupon the investigational product dosing may resume. For patients with screening eGFR ≥60 mL/min/1.73 m², when the subsequent eGFR falls to <40 mL/min/1.73 m², investigational product will be withheld until their eGFR becomes ≥50 mL/min/1.73 m², whereupon the investigational product dosing may resume (see Section 8.1.1).

## 7.3. Blinding

This is a double-blind study. To preserve the blinding of the study, a minimum number of Lilly personnel will see the randomization table and treatment assignments before the study is complete. All study assessments will be performed by study personnel who are blinded to the patient's treatment group. Except in clinical circumstances where unblinding is required, the patients, investigators, Lilly study team, and any personnel interacting directly with patients or investigative sites will remain blinded to baricitinib and placebo assignment until after completion of the Double-Blinded Treatment Period. It is expected that the need for unblinding a patient's treatment prior to completion of the Double-Blinded Treatment Period will be extremely rare. Every effort should be made to preserve the blind unless there is a compelling reason that knowledge of the specific treatment would alter the medical care of the patient. In case of an emergency, the investigator has the sole responsibility for determining if unblinding of a patient's treatment assignment is warranted for medical management of the event. Patient safety must always be the first consideration in making such a determination. If a patient's treatment assignment is unblinded, Lilly must be notified immediately. If the investigator decides that unblinding is warranted, it is the responsibility of the investigator to promptly document the decision and rationale and notify Lilly as soon as possible.

Emergency unblinding for AEs may be performed through the IWRS. This option may be used ONLY if the patient's well-being requires knowledge of the patient's treatment assignment. All unblinding events are recorded and reported by the IWRS. If an investigator, site personnel performing assessments, or patient is unblinded, the patient must be discontinued from the study. In cases where there are ethical reasons to have the patient remain in the study, the investigator must obtain specific approval from a Lilly clinical research physician for the patient to continue in the study.

Processes to maintain blinding during the interim analysis conducted by the DMC are described in Section 10.3.7.1.

# 7.4. Dosage Modification

Not applicable.

## 7.5. Preparation/Handling/Storage/Accountability

All investigational product (used and partially used) will be returned to the sponsor or destroyed at site level with the sponsor's written approval. In some cases, sites may destroy the material if, during the investigative site selection, the evaluator has verified and documented that the site has appropriate facilities and written procedures to dispose of clinical trial materials.

Follow storage and handling instructions on the investigational product packaging.

## 7.6. Treatment Compliance

Patient compliance with study medication will be assessed at each visit during the treatment period (Visit 3 through Visit 8) by counting returned tablets.

A patient will be considered significantly noncompliant if he or she misses more than 20% of the prescribed doses of investigational product during the study, unless the patient's investigational product is withheld by the investigator for safety reasons. Similarly, a patient will be considered significantly noncompliant if he or she is judged by the investigator to have intentionally or repeatedly taken 20% more than the prescribed amount of medication during the study.

Patients will be counseled by study staff on the importance of taking the investigational product as prescribed, as appropriate.

Patients' compliance will be further defined in the statistical analysis plan (SAP).

## 7.7. Concomitant Therapy

All concomitant medication, whether prescription or over the counter, used at baseline and/or during the course of the study, must be recorded on the Concomitant Medication electronic case report form (eCRF). Patients will be instructed to consult the investigator or other appropriate study personnel at the site before taking any new medications or supplements during the study. For AD therapies permitted as part of rescue therapy, see Section 7.7.3.

#### 7.7.1. Prohibited Medications and Procedures

# **Prohibited Medications and Procedures Not Requiring Interruption of Investigational Product**

The following therapies will not be allowed during the course of the study and, if taken by or administered to the patient, the prohibited therapy must be discontinued.

- TCS, TCNIs (e.g., tacrolimus and pimecrolimus), or topical PDE 4 inhibitor (i.e., crisaborole) except when given as rescue therapy as described in Section 7.7.3.
- topical antihistamines or sedating, systemic antihistamines including, but not limited to, alimemazine, chlorphenamine, clemastine, cyproheptadine, diphenhydramine, hydroxyzine, ketotifen, and promethazine
- leukotriene inhibitors (e.g., montelukast [Singulair], zafirlukast [Accolate], and zileuton [Zyflo])
- allergen immunotherapy

- phototherapy including PUVA (psoralen and ultraviolet A), ultraviolet B, tanning booth and excimer laser
- bleach baths

#### **Prohibited Medications Requiring Temporary Interruption of Investigational Product**

The following therapies will not be allowed during the course of the study and, if taken by or administered to the patient, temporary interruption of investigational product is required.

- live vaccines (including Bacillus Calmette-Guérin [BCG] or herpes zoster), (see Exclusion Criterion [27])
  - o For BCG vaccination, investigational product should be temporarily interrupted for 12 weeks.
  - For herpes zoster vaccination, investigational product should be temporarily interrupted for 4 weeks.
- probenecid: if a patient is inadvertently started on probenecid, IP should be temporarily interrupted, and can be resumed after patient has discontinued probenecid. If a patient is not able to discontinue probenecid, then IP should be permanently discontinued

#### **Prohibited Medications Requiring Permanent Discontinuation of Investigational Product**

- systemic corticosteroids
- any systemic therapy, investigational or commercial (approved or off label use), used for the treatment of AD or symptoms of AD (except for antihistamines, as specified above)
- other JAK inhibitors (e.g., tofacitinib and ruxolitinib)
- systemic immunosuppressive/immunomodulatory substances, including, but not limited to, cyclosporine, methotrexate, mycophenolate mofetil, interferon  $\gamma$ , azathioprine, or biologic agents

Note: In the event that these prohibited medications were inadvertently used, agreement and documentation to continue investigational product must be sought from sponsor.

#### 7.7.2. Permitted Medications and Procedures

Treatment with concomitant AD therapies during the study is permitted only as described below.

- Daily use of emollients is required as background treatment. Moisturizers with additives such as antiprurities or antiseptics are not permitted. If daily applications are missed, it will not be considered a protocol violation.
  - o Patients should not apply emollients on the day of their study visit prior to the procedures to allow adequate assessment of skin dryness.
- For those patients on stable dosing of prescription sleep medications at entry, downward dose adjustments or discontinuation of treatment may occur during the study.

- Nonsedating antihistamines including, but not limited to, acrivastine, bilastine, cetirizine, desloratadin, fexofenadine, levocetirizine, loratadine, mizolastine, and rupatadine are allowed.
- Single intra-articular or soft tissue (bursa, tendons, and ligaments) corticosteroid injection is allowed during the 16-week double-blind, placebo-controlled period.
- Intranasal or inhaled steroid use is allowed.
- Topical anesthetics and topical and systemic anti-infective medications are allowed.
- Nonlive seasonal vaccinations and/or emergency vaccination, such as rabies or tetanus vaccinations, are allowed.

Any changes of these concomitant medications must be recorded in the Concomitant Therapy of Special Interest eCRF.

Treatment with concomitant therapies for other medical conditions such as diabetes and hypertension is permitted during the study.

## 7.7.3. Rescue Therapy

#### Criteria for rescue therapy initiation

Investigators should attempt to manage patients with emollients, however, investigators are allowed to rescue patients who are experiencing unacceptable or worsening symptoms of AD at any time. Prior to rescue, it is recommended that increased frequency of emollient use is attempted to at least twice a day or more in an effort to control symptoms. The rationale for rescue will be documented.

#### Choice of rescue therapy treatment

- Triamcinolone 0.1% cream and/or hydrocortisone 2.5% ointment. Where possible, both of these treatments will be supplied by the sponsor. In the event where providing 1 or both of these topical formulations is not possible, an alternate, equivalent potency TCS cream and/or ointment may be provided by the sponsor. TCS use, supplied by the sponsor, should be recorded via weight of returned tubes as indicated in the Schedule of Activities (Section 2).
  - o In the event that the sponsor is unable to supply TCS, commercially available triamcinolone 0.1% cream and/or hydrocortisone 2.5% ointment may be supplied by the sites. Where providing triamcinolone 0.1% cream and/or hydrocortisone 2.5% ointment is not possible, an equivalent-potency TCS cream and/or ointment that is in line with local practices can be supplied. Refer to Appendix 7 for guidance on potency equivalence.
  - If the TSC supplied by the sponsor is not considered suitable for an individual patient, an equivalent-potency TCS cream and/or ointment that is in line with

local practices can be supplied by the sites. Refer to Appendix 7 for guidance on potency equivalence.

- Investigators may also select to use TCNIs and/or crisaborole where approved, although use of either during the study is neither encouraged nor provided. If TCNIs are prescribed, use should be limited to problem areas only (e.g., face, neck, skin folds, genital areas, etc.).
- On the days of study visits, topical therapy should not be applied before the patient has undergone all study procedures and clinical evaluations in order to allow adequate assessment of skin dryness
- Patients rescued to topical therapy will continue to take investigational product and use of rescue therapy will be documented in the eCRF.

In patients who do not improve sufficiently with the provided rescue topical therapy after 7 days, a higher potency TCS may be used (see Appendix 7) and investigational product may continue. Higher potency TCS will not be supplied centrally by the sponsor. It is recommended that if a patient reaches "clear" to "almost clear" skin after topical rescue, then medium- and/or high-potency TCS and TCNI should be stopped, and low–potency TCS (e.g., hydrocortisone 2.5% ointment) should be used once daily for an additional 7 days, then stopped. If lesions return, patients can be retreated with TCS with or without TCNIs and/or crisaborole as before at the discretion of the investigator.

If topical rescue therapy as described above fails to sufficiently control AD symptoms, then oral systemic medications may be used as rescue (e.g., corticosteroids, cyclosporine, methotrexate); however, investigational product will be required to be permanently discontinued for the remainder of the 16-week study duration. If these medications are needed for other medical conditions (e.g., asthma flare), they will still be treated as rescue medications. These patients are still eligible to enter the long-term extension study (JAHN), if they complete the schedule of study visits through Visit 8 (Week 16) and are also able to complete a minimum 4-week washout from oral systemic rescue medications (which can occur during the screening period for Study JAHN).

Investigators should make every attempt to conduct efficacy and safety assessments immediately before administering any rescue treatment. An unscheduled visit can be used for this purpose if necessary.

# 7.8. Treatment after the End of the Study

# 7.8.1. Study Extensions

Patients who complete this study through Visit 8 may be eligible to participate in Study JAHN, if enrollment criteria for Study JAHN are met.

## 7.8.2. Continued Access

After the conclusion of the study, continued access to baricitinib will not be provided to patients who are not eligible for or who do not choose to participate in Study JAHN. Patients will be referred to their local treatment centers for AD therapy as clinically indicated.

## 8. Discontinuation Criteria

## 8.1. Discontinuation from Study Treatment

## 8.1.1. Temporary Interruption from Investigational Product

In some circumstances, it may be necessary to temporarily interrupt treatment as a result of AEs or abnormal laboratory values that may have an unclear relationship to investigational product. For example, investigational product should be temporarily interrupted if the patient experiences a cardiovascular adverse event considered to be related to study treatment, is graded as moderate (Grade 2 according to Common Terminology Criteria for Adverse Events [CTCAE] Version 3.0), and that does not resolve promptly with supportive care. Except in cases of emergency, it is recommended that the investigator consult with Lilly (or its designee) before temporarily interrupting therapy for reasons other than those defined in Table JAHL.4.

For the abnormal laboratory findings and clinical events (regardless of relatedness) listed in Table JAHL.4, specific guidance is provided for temporarily interrupting treatment and when treatment may be restarted. Retest frequency and timing of follow-up laboratory tests to monitor the abnormal finding is at the discretion of the investigator. Investigational product that was temporarily interrupted because of an AE or abnormal laboratory value not specifically covered in Table JAHL.4 may be restarted at the discretion of the investigator.

Table JAHL.4. Criteria for Temporary Interruption of Investigational Product

| Hold Investigational Product if the Following<br>Laboratory Test Results or Clinical Events Occur: | Investigational Product May Be Resumed When: |
|---|---|
| WBC count <2000 cells/μL | WBC count ≥2500 cells/μL |
| $(<2.00x10^3/\mu L \text{ or } <2.00 \text{ GI/L})$ | $(\ge 2.50 \times 10^3 / \mu L \text{ or } \ge 2.50 \text{ GI/L})$ |
| ANC <1000 cells/μL | ANC ≥1200 cells/μL |
| $(<1.00 \times 10^3/\mu L \text{ or } <1.00 \text{ GI/L})$ | $(\ge 1.20 \times 10^3 / \mu L \text{ or } \ge 1.20 \text{ GI/L})$ |
| Lymphocyte count <500 cells/μL | Lymphocyte count ≥750 cells/μL |
| $(<0.50x10^3/\mu L \text{ or } <0.50 \text{ GI/L})$ | $(\ge 0.75 \times 10^3 / \mu L \text{ or } \ge 0.75 \text{ GI/L})$ |
| Platelet count <75,000/μL | Platelet count ≥100,000/μL |
| $(<75x10^3/\mu L \text{ or } <75 \text{ GI/L})$ | $(\geq 100 \times 10^3 / \mu L \text{ or } \geq 100 \text{ GI/L})$ |
| eGFR <40 mL/min/1.73 m <sup>2</sup> (from serum creatinine) for | eGFR ≥50 mL/min/1.73 m <sup>2</sup> |
| patients with screening eGFR ≥60 mL/min/1.73 m <sup>2</sup> | |
| eGFR <30 mL/min/1.73 m <sup>2</sup> (from serum creatinine) for | eGFR ≥40 mL/min/1.73 m <sup>2</sup> |
| patients with screening eGFR ≥40 to <60 mL/min/1.73 m <sup>2</sup> | |
| ALT or AST >5x ULN | ALT and AST return to <2x ULN, and IP is not |
| | considered to be the cause of enzyme elevation |
| Hemoglobin <8 g/dL (<80.0 g/L) | Hemoglobin ≥10 g/dL (≥100.0 g/L) |
| Symptomatic herpes zoster | All skin lesions have crusted and are resolving |
| Infection that, in the opinion of the investigator, merits the | Resolution of infection |
| IP being interrupted | |
| Clinical features of VTE (such as deep vein thrombosis or | After evaluation and institution of appropriate |
| pulmonary embolism) are present <sup>a</sup> | treatment of VTEb |

Abbreviations: ALT = alanine aminotransferase; ANC = absolute neutrophil count; AST = aspartate aminotransferase; eGFR = estimated glomerular filtration rate; IP = investigational product; ULN = upper limit of normal; VTE = venous thromboembolic event; WBC = white blood cell.

- <sup>a</sup> Evaluate promptly and institute appropriate treatment. If upon evaluation VTE is ruled out and no other temporary or permanent discontinuation criteria are met, then IP may be resumed.
- b If after evaluation and institution of treatment the investigator deems that the patient is still at significant risk, or if this would constitute a second VTE for the patient, then IP should be discontinued permanently

Although temporary interruption of investigational product is not a requirement at times of increased potential risk of VTE (e.g., surgery, significant air travel, or other situations involving prolonged immobilization) we recommend following appropriate VTE prophylaxis guidelines to help manage the VTE risk under these circumstances.

For specific guidance on temporary interruption of IP after use of a prohibited medication, please refer to Section 7.7.1 (Prohibited Medications and Procedures).

Lastly, investigational product should be temporarily interrupted for suicidal ideation or any suicide-related behaviors as assessed by the following patient responses on the C-SSRS:

- A "yes" answer to Question 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) or
- A "yes" answer to Question 5 (Active Suicidal Ideation with Specific Plan and Intent) on the "Suicidal Ideation" portion of the C-SSRS or
- A "yes" answer to any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act or behavior) on the "Suicidal Behavior" portion of the C-SSRS.

NOTE: Prior to resumption of investigational product, it is recommended that a patient be assessed by a psychiatrist or appropriately trained professional to assist in deciding whether the subject should remain on investigational product and ultimately continued participation in the study. A patient does not necessarily have to have investigational product interrupted if they have self-injurious behavior that would be classified as non-suicidal self-injurious behavior.

# 8.1.2. Permanent Discontinuation from Investigational Product

Investigational product should be permanently discontinued if the patient requests to discontinue investigational product.

Discontinuation of the investigational product for abnormal liver tests should be considered by the investigator when a patient meets 1 of the following conditions after consultation with the Lilly-designated medical monitor:

- ALT or AST >8x ULN
- ALT or AST >5x ULN for more than 2 weeks
- ALT or AST >3x ULN and total bilirubin level (TBL) >2x ULN or international normalized ratio (INR) >1.5

- ALT or AST >3x ULN with the appearance of fatigue, nausea, vomiting, right upper-quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%)
- ALP >3x ULN
- ALP >2.5x ULN and TBL >2x ULN
- ALP >2.5x ULN with the appearance of fatigue, nausea, vomiting, right quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%)

**NOTE:** Patients who are discontinued from investigational product due to a hepatic event or liver test abnormality should have additional hepatic safety data collected via the hepatic safety eCRF.

Investigational product should be permanently discontinued if any of the following laboratory abnormalities are observed:

- white blood cell count <1000 cells/ $\mu$ L (1.00x10<sup>3</sup>/ $\mu$ L or 1.00 GI/L)
- ANC  $<500 \text{ cells/}\mu\text{L} (0.50 \times 10^3/\mu\text{L} \text{ or } 0.50 \text{ GI/L})$
- lymphocyte count  $<200 \text{ cells/}\mu\text{L}$  (0.20x10<sup>3</sup>/ $\mu\text{L}$  or 0.20 GI/L)
- hemoglobin <6.5 g/dL (<65.0 g/L).

NOTE: Temporary interruption rules (see Section 8.1.1) must be followed where applicable. For laboratory values that meet permanent discontinuation thresholds, investigational product should be discontinued. However, if in the opinion of the investigator the laboratory abnormality is due to intercurrent illness such as cholelithiasis or another identified factor, laboratory tests may be repeated. Only when the laboratory value meets resumption thresholds (Table JAHL.4) following the resolution of the intercurrent illness or other identified factor, may the investigator restart investigational product, after consultation with the Lilly-designated medical monitor.

In addition, patients will be discontinued from investigational product in the following circumstances:

- pregnancy
- malignancy (except for successfully treated basal or squamous cell skin carcinoma)
- hepatitis B virus DNA is detected with a value above limit of quantitation or 2 sequential tests return a value of below the limit of quantitation (see Section 9.4.8).
- develop a second VTE
- certain prohibited medications are taken per Section 7.7.1 (Prohibited Medications and Procedures).

If a patient discontinues investigational product for any reason, the patient is encouraged to remain in the study through Week 16 (Visit 8) and follow the regular visit schedule to provide

the primary efficacy and safety data. Patients discontinuing from the investigational product prematurely for any reason should complete AE and other follow-up procedures per Section 2 (Schedule of Activities), Section 9.2 (Adverse Events), and Section 9.4 (Safety) of this protocol.

## 8.1.3. Discontinuation of Inadvertently Enrolled Patients

If the sponsor or investigator identifies a patient who did not meet enrollment criteria and was inadvertently enrolled, then the patient should be discontinued from study treatment unless there are extenuating circumstances that make it medically necessary for the patient to continue on study treatment. If the investigator and the sponsor clinical research physician agree it is medically appropriate to continue, the investigator must obtain documented approval from the sponsor clinical research physician to allow the inadvertently enrolled patient to continue in the study with or without treatment with investigational product. Safety follow up is as outlined in Section 2 (Schedule of Activities), Section 9.2 (Adverse Events), and Section 9.4 (Safety) of this protocol.

## 8.2. Discontinuation from the Study

Patients may choose to withdraw from the study for any reason at any time, and the reason for early withdrawal will be documented.

Some possible reasons that may lead to permanent discontinuation include the following:

- enrollment in any other clinical study involving an investigational product or enrollment in any other type of medical research judged not to be scientifically or medically compatible with this study.
- participation in the study needs to be stopped for medical, safety, regulatory, or other reasons consistent with applicable laws, regulations, and good clinical practice (GCP).
- investigator decision
  - The investigator decides that the patient should be discontinued from the study.
  - O If the patient, for any reason, requires treatment with another therapeutic agent (not allowed as part of rescue therapy [Section 7.7.3]) that has been demonstrated to be effective for treatment of the study indication, discontinuation from the study occurs prior to introduction of the new agent.
- patient decision
  - The patient requests to be withdrawn from the study.

Patients discontinuing from the study prematurely for any reason should complete AE and other safety follow-up per Section 2 (Schedule of Activities), Section 9.2 (Adverse Events), and Section 9.4 (Safety) of this protocol.

# 8.3. Lost to Follow-Up

A patient will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site. Site personnel are expected to make diligent attempts to contact patients who fail to return for a scheduled visit or were otherwise unable to be followed up by the site.

# 9. Study Assessments and Procedures

Section 2 lists the Schedule of Activities, with the study procedures and their timing (including tolerance limits for timing).

Appendix 2 and Appendix 4 list the laboratory tests that will be performed for this study.

Unless otherwise stated in the subsections below, all samples collected for specified laboratory tests will be destroyed within 60 days of receipt of confirmed test results. Certain samples may be retained for a longer period, if necessary, to comply with applicable laws, regulations, or laboratory certification standards.

## 9.1. Efficacy Assessments

## 9.1.1. Primary Efficacy Assessments

**Validated Investigator's Global Assessment for Atopic Dermatitis (vIGA-AD):** The IGA used in this study, the vIGA-AD (referred to as the IGA throughout the protocol) measures the investigator's global assessment of the patient's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.

## 9.1.2. Secondary Efficacy Assessments

## 9.1.2.1. Eczema Area and Severity Index Scores

The EASI assesses extent of disease at 4 body regions and measures 4 clinical signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3. The EASI confers a maximum score of 72. The EASI evaluates 2 dimensions of AD: disease extent and clinical signs (Hanifin et al. 2001).

Body surface area affected by AD will be derived from data collected as part of the EASI assessment.

## 9.1.2.2. SCORing Atopic Dermatitis

The SCORing Atopic Dermatitis (SCORAD) index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness. The SCORAD index also assesses subjective symptoms of pruritus and sleep loss. These 3 aspects: extent of disease, disease severity, and subjective symptoms combine to give a maximum possible score of 103 (Stalder et al. 1993; Kunz et al. 1997; Schram et al. 2012).

#### 9.1.2.3. Hospital Anxiety Depression Scale

The Hospital Anxiety Depression Scale (HADS) is a 14-item self-assessment scale that determines the levels of anxiety and depression that a patient is experiencing over the past week. The HADS utilizes a 4-point Likert scale (e.g., 0 to 3) for each question and is intended for ages 12 to 65 years (Zigmond and Snaith 1983; White et al. 1999). Scores for each domain (anxiety

and depression) can range from 0 to 21, with higher scores indicating greater anxiety or depression (Zigmond and Snaith 1983; Snaith 2003).

## 9.1.3. Health Outcomes and Quality-of-Life Measures

The patient self-reported questionnaires will be administered via either an electronic patient diary or via an electronic tablet and in countries where the questionnaires have been translated into the native language of the region and linguistically validated.

#### 9.1.3.1. Patient-Oriented Eczema Measure

The POEM is a simple, 7-item, patient-administered scale that assesses disease severity in children and adults. Patients respond to questions about the frequency of 7 symptoms (itching, sleep disturbance, bleeding, weeping/oozing, cracking, flaking, and dryness/roughness) over the last week. Response categories include "No days," "1-2 days," "3-4 days," "5-6 days," and "Every day" with corresponding scores of 0, 1, 2, 3, and 4, respectively. Scores range from 0-28 with higher total scores indicating greater disease severity (Charman et al. 2004).

#### 9.1.3.2. Itch Numeric Rating Scale

The Itch Numeric Rating Scale (NRS) is a patient-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a patient's itching is indicated by selecting the number that best describes the worst level of itching in the past 24 hours (Naegeli et al. 2015; Kimball et al. 2016).

#### 9.1.3.3. Nocturnal Sleep-Wake and Itch Patterns

An actigraphy device, a hypoallergenic device worn on the wrist, will be used to collect sleep-wake patterns and quantify nocturnal scratching events. Each patient will be dispensed 2 actigraphy devices. One will be worn on the wrist at all times and the other will be worn only during hours of sleep (one on each wrist). Further details on use of the device will be provided in other instructional materials.

#### 9.1.3.4. Atopic Dermatitis Sleep Scale

The Atopic Dermatitis Sleep Scale (ADSS) is a 3-item, patient-administered questionnaire developed to assess the impact of itch on sleep including difficulty falling asleep, frequency of waking, and difficulty getting back to sleep last night. Patient's rate their difficulty falling asleep and difficulty getting back to sleep, items 1 and 3, respectively, using a 5-point Likert-type scale with response options ranging from 0 "not at all" to 4 "very difficult." Patients report their frequency of waking last night, item 2, by selecting the number of times they woke up each night, ranging from 0 to 29 times. The ADSS is designed to be completed each day with respondents thinking about sleep "last night." Each item is scored individually.

## 9.1.3.5. Skin Pain Numeric Rating Scale

Skin Pain NRS is a patient-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no pain" and 10 representing "worst pain imaginable." Overall severity of a patient's skin pain is indicated by selecting the number that best describes the worst level of skin pain in the past 24 hours.

#### 9.1.3.6. Patient Global Impression of Severity

The Patient Global Impression of Severity–Atopic Dermatitis (PGI-S-AD) is a single-item question asking the patient how they would rate their overall AD symptoms over the past 24 hours. The 5 categories of responses range from "no symptoms" to "severe."

#### 9.1.3.7. Dermatology Life Quality Index

The Dermatology Life Quality Index (DLQI) is a simple, patient-administered, 10-item, validated, quality-of-life questionnaire that covers 6 domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The recall period of this scale is over the "last week." Response categories include "not at all," "a lot," and "very much," with corresponding scores of 1, 2, and 3, respectively, and unanswered ("not relevant") responses scored as 0. Scores range from 0-30 with higher scores indicating greater impairment of quality of life. A DLQI total score of 0 to 1 is considered as having no effect on a patient's health-related QoL (Hongbo et al. 2005), and a 4-point change from baseline is considered as the minimal clinically important difference threshold (Khilji et al. 2002; Basra et al. 2015).

#### 9.1.3.8. European Quality of Life-5 Dimensions-5 Levels

The European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) is a standardized measure of health status that provides a simple, generic measure of health for clinical and economic appraisal. The EQ-5D-5L consists of 2 components: a descriptive system of the respondent's health and a rating of his or her current health state using a 0 to 100 mm VAS. The descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The respondent is asked to indicate his or her health state by ticking (or placing a cross) in the box associated with the most appropriate statement in each of the 5 dimensions. It should be noted that the numerals 1 to 5 have no arithmetic properties and should not be used as an ordinal score. The VAS records the respondent's self-rated health on a vertical VAS where the endpoints are labeled "best imaginable health state" and "worst imaginable health state." This information can be used as a quantitative measure of health outcome. The EQ-5D-5L health states, defined by the EQ-5D-5L descriptive system, may be converted into a single summary index by applying a formula that essentially attaches values (also called weights) to each of the levels in each dimension (Herdman et al. 2011; EuroQol Group 2015 [WWW]).

# 9.1.3.9. Work Productivity and Activity Impairment Questionnaire-Atopic Dermatitis

The Work Productivity and Activity Impairment Questionnaire—Atopic Dermatitis (WPAI-AD) records impairment due to AD during the past 7 days. The WPAI-AD consists of 6 items grouped into 4 domains: absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity impairment. Scores are calculated as impairment percentages (Reilly et al. 1993), with higher scores indicating greater impairment and less productivity.

## 9.1.4. Appropriateness of Assessments

All assessments utilized in this study are standard, widely used, and generally recognized as reliable, accurate, and relevant except ADSS and Skin Pain NRS, which are currently being developed and validated according to regulatory guidances.

#### 9.2. Adverse Events

Investigators are responsible for monitoring the safety of patients who have entered this study and for alerting Lilly or its designee to any event that seems unusual, even if this event may be considered an unanticipated benefit to the patient.

The investigator is responsible for the appropriate medical care of patients during the study.

Investigators must document their review of each laboratory safety report.

The investigator remains responsible for following, through an appropriate health care option, AEs that are serious or otherwise medically important, considered related to the investigational product or the study, or that caused the patient to discontinue the investigational product before completing the study. The patient should be followed until the event resolves, stabilizes with appropriate diagnostic evaluation, or is reasonably explained. The frequency of follow-up evaluations of the AE is left to the discretion of the investigator.

Lack of drug effect is not an AE in clinical studies, because the purpose of the clinical study is to establish treatment effect.

After the ICF is signed, study site personnel will record via eCRF the occurrence and nature of each patient's preexisting conditions, including clinically significant signs and symptoms of the disease under treatment in the study. In addition, site personnel will record any change in the condition(s) and any new conditions as AEs. Investigators should record their assessment of the potential relatedness of each AE to investigational product, via eCRF.

The investigator will interpret and document whether or not an AE has a reasonable possibility of being related to study treatment, study device, or a study procedure, taking into account the disease, concomitant treatment, or pathologies. A "reasonable possibility" means that there is a cause-and-effect relationship between the investigational product, study device, and/or study procedure and the AE. The investigator answers yes/no when making this assessment.

Planned surgeries and nonsurgical interventions should not be reported as AEs unless the underlying medical condition has worsened during the course of the study.

If a patient's investigational product is discontinued as a result of an AE, study site personnel must report this to Lilly or its designee via eCRF, clarifying if possible the circumstances leading to any dosage modifications, or discontinuations of treatment.

#### 9.2.1. Serious Adverse Events

An SAE is any AE from this study that results in 1 of the following outcomes:

death

- initial or prolonged inpatient hospitalization
- a life-threatening experience (i.e., immediate risk of dying)
- persistent or significant disability/incapacity
- congenital anomaly/birth defect
- important medical events that may not be immediately life threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent 1 of the other outcomes listed in the definition above. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

All AEs occurring after signing the ICF are recorded in the eCRF and assessed for serious criteria. The SAE reporting to the sponsor begins after the patient has signed the ICF and has received investigational product. However, if an SAE occurs after signing the ICF, but prior to receiving investigational product, the SAE should be reported to the sponsor as per SAE reporting requirements and timelines if it is considered reasonably possibly related to study procedure.

Study site personnel must alert Lilly or its designee of any SAE within 24 hours of investigator awareness of the event via a sponsor-approved method. If alerts are issued via telephone, they are to be immediately followed with official notification on study-specific SAE forms. This 24-hour notification requirement refers to the initial SAE information and all follow-up SAE information. Patients with a serious hepatic AE should have additional data collected using the hepatic safety eCRF.

Pregnancy (during maternal or paternal exposure to investigational product) does not meet the definition of an AE. However, to fulfill regulatory requirements, any pregnancy should be reported following the SAE process to collect data on the outcome for both mother and fetus.

Investigators are not obligated to actively seek AEs or SAEs in subjects once they have discontinued and/or completed the study (the patient summary CRF has been completed). However, if the investigator learns of any SAE, including a death, at any time after a subject has been discharged from the study, and he or she considers the event reasonably possibly related to the study treatment or study participation, the investigator must promptly notify Lilly.

## 9.2.1.1. Suspected Unexpected Serious Adverse Reactions

Suspected unexpected serious adverse reactions (SUSARs) are serious events that are not listed in the IB and that the investigator identifies as related to investigational product or procedure. United States 21 CFR 312.32 and European Union Clinical Trial Directive 2001/20/EC and the associated detailed guidances or national regulatory requirements in participating countries require the reporting of SUSARs. Lilly has procedures that will be followed for the recording and expedited reporting of SUSARs that are consistent with global regulations and the associated detailed guidances.

## 9.2.2. Adverse Events of Special Interest

Adverse events of special interest will include the following:

- infections (including TB, herpes zoster, or opportunistic infections)
- malignancies
- hepatic events (see Section 9.4.9)
- major adverse cardiovascular events (MACE) (see Section 9.4.10)
- thrombotic events (such as deep vein thrombosis [DVT] and pulmonary embolism).

Sites will provide details on these AEs as instructed on the eCRF and may be asked for additional description by Lilly.

## 9.2.3. Complaint Handling

Lilly collects product complaints on investigational products and drug delivery systems used in clinical studies to ensure the safety of study participants, monitor quality, and to facilitate process and product improvements.

Patients will be instructed to contact the investigator as soon as possible if he or she has a complaint or problem with the investigational product so that the situation can be assessed.

#### 9.3. Treatment of Overdose

Refer to the IB.

# 9.4. Safety

Any clinically significant findings from ECG testing, physical examination, vital signs measurements, or laboratory measurements that result in a diagnosis and that occur after the patient receives the first dose of study treatment should be reported to Lilly or its designee as an AE via eCRF.

# 9.4.1. Electrocardiograms

A single 12-lead standard ECG will be obtained locally at Visit 1 and read by a qualified physician (the investigator or qualified designee) at the site to determine whether the patient meets entry criteria.

Electrocardiograms may be obtained at additional times, when deemed clinically necessary.

# 9.4.2. Vital Signs

For each patient, vital signs should be measured according to the Schedule of Activities (Section 2).

## 9.4.3. Physical Exam

For each patient, a complete physical examination (excluding pelvic and rectal examinations) will be performed at Visit 1 (Screening). A symptom-directed physical examination will be performed at other visits as specified in the Schedule of Activities (Section 2). A complete physical examination may be repeated at the investigator's discretion at any time a patient presents with physical complaints.

## 9.4.4. Laboratory Tests

For each patient, laboratory tests detailed in Appendix 2 should be conducted according to the Schedule of Activities (Section 2). With the exception of laboratory test results that may unblind the study, Lilly or its designee will provide the investigator with the results of laboratory tests analyzed by a central vendor, if a central vendor is used for the clinical trial.

## 9.4.5. Columbia Suicide Severity Rating Scale

The C-SSRS captures the occurrence, severity, and frequency of suicidal ideation and/or behavior during the assessment period. The scale includes suggested questions to solicit the type of information needed to determine if suicidal ideation and/or behavior occurred. The C-SSRS is administered by an appropriately trained health care professional with at least 1 year of patient care/clinical experience. The tool was developed by the National Institute of Mental Health trial group for the purpose of being a counterpart to the Columbia Classification Algorithm of Suicide Assessment categorization of suicidal events. For this study, the scale has been adapted (with permission from the scale authors) to include only the portion of the scale that captures the occurrence of the 11 preferred ideation and behavior categories.

The nonleading AE collection should occur prior to the collection of the C-SSRS. If a suicide-related event is discovered *during the C-SSRS* but was not captured during the nonleading AE collection, sites should not change the AE form. If an event is serious or leads to discontinuation, this is an exception where the SAE and/or AE leading to discontinuation should be included on the AE form and the process for reporting SAEs should be followed.

# 9.4.6. Self-Harm and Follow-up Supplement Forms

Suicide-related events (behavior and/or ideations) will be assessed and evaluated at every visit with the administration of the C-SSRS and the Self-Harm Supplement Form. The Self-Harm Supplement Form is a single question to enter the number of suicidal behavior events, possible suicide behaviors, or nonsuicidal self-injurious behaviors. If the number of behavioral events is greater than zero, it will lead to the completion of the self-harm follow-up form. The self-harm follow-up form is a series of questions that provides a more detailed description of the behavior cases.

# 9.4.7. Chest x-ray and Tuberculosis Testing

A posterior—anterior view chest x-ray will be obtained locally at screening (Visit 1), unless results from a chest x-ray obtained within 6 months prior to the study are available. The chest x-ray will be reviewed by the investigator or his or her designee to exclude patients with active

TB infection. In addition, patients will be tested at screening (Visit 1) for evidence of active or latent TB as described in the exclusion criteria, Section 6.2.

Investigators should follow local guidelines for monitoring patients for TB if a patient is at high risk for acquiring TB or reactivation of latent TB.

## 9.4.8. Hepatitis B Virus DNA Monitoring

Patients who are HBcAb positive and HBV DNA negative (undetectable) at Visit 1 will require measurement of HBV DNA at Week 16 (Visit 8) or early termination visit, regardless of their hepatitis B surface antibody (HBsAb) status.

The following actions should be taken in response to HBV DNA test results:

- If a single result is obtained with a value "below limit of quantitation," the test should be repeated within approximately 2 weeks. If the repeat test result is "target not detected," monitoring will resume for those patients enrolling in the long-term extension study, JAHN.
- If the patient has 2 or more test results with a value "below limit of quantitation" or a test result above the limit of quantitation, the patient will be permanently discontinued from investigational product (see Section 8.1.2) and should be referred to a hepatology specialist.

## 9.4.9. Hepatic Safety Monitoring and Data Collection

If a study patient experiences elevated ALT  $\ge 3x$  ULN, ALP  $\ge 2x$  ULN, or elevated TBL  $\ge 2x$  ULN, liver testing (Appendix 4) should be repeated within 3 to 5 days including ALT, AST, ALP, TBL, direct bilirubin, gamma-glutamyl transferase, and creatine kinase to confirm the abnormality and to determine if it is increasing or decreasing. If the abnormality persists or worsens, clinical and laboratory monitoring should be initiated by the investigator and in consultation with the study medical monitor. Monitoring of ALT, AST, TBL, and ALP should continue until levels normalize or return to approximate baseline levels.

Discontinuation criteria of investigational products, either temporary interruption or permanent discontinuation, due to abnormal ALT, AST, TBL, or ALP, are detailed in Section 8.1.

Additional safety data should be collected via the hepatic eCRF if 1 or more of the following conditions occur:

- elevation of serum ALT to ≥5x ULN on 2 or more consecutive blood tests
- elevated serum TBL to  $\geq 2x$  ULN (except for cases of known Gilbert's syndrome)
- elevation of serum ALP to  $\ge 2x$  ULN on 2 or more consecutive blood tests
- patient discontinued from treatment due to a hepatic event or abnormality of liver tests
- hepatic event considered to be an SAE.

See Appendix 4 and Appendix 5 for a description of hepatic laboratory values that warrant exclusion from the study, temporary or permanent discontinuation of investigational product, or additional safety collection via the hepatic eCRF.

## 9.4.10. Safety Monitoring

Lilly will periodically review evolving aggregate safety data within the study by appropriate methods.

In the event that safety monitoring uncovers an issue that needs to be addressed by unblinding at the group level, only members of the DMC (an advisory group for this study formed to protect the integrity of data [refer to Interim Analyses section, Section 10.3.7]) can conduct additional analyses of the safety data.

The Lilly clinical research physician will monitor safety data throughout the course of the study. Lilly will review SAEs within time frames mandated by company procedures. The Lilly clinical research physician will, as is appropriate, consult with the functionally independent Global Patient Safety therapeutic area physician or clinical scientist and periodically review trends in safety data and laboratory analytes. Any concerning trends in frequency or severity noted by an investigator and/or Lilly (or designee) may require further evaluation.

All deaths and SAE reports will be reviewed in a blinded manner by Lilly during the clinical trial. These reports will be reviewed to ensure completeness and accuracy but will not be unblinded to Lilly during the clinical trial. If a death or a clinical AE is deemed serious, unexpected, and possibly related to investigational product, only Lilly Global Patient Safety will be unblinded for regulatory reporting and safety monitoring purposes. These measures will preserve the integrity of the data collected during this trial and minimize any potential for bias while providing for appropriate safety monitoring.

Investigators will monitor vital signs and carefully review findings that may be associated with cardiovascular and venous thrombotic events. Adverse event reports and vital signs will be collected at each study visit. The cardiovascular monitoring plan includes the following:

- regular monitoring of lipid levels
- potential MACE (cardiovascular death, MI, stroke), other cardiovascular events (such as hospitalization for unstable angina, hospitalization for heart failure, serious arrhythmia, resuscitated sudden death, cardiogenic shock, coronary revascularization such as coronary artery bypass graft or percutaneous coronary intervention), venous thrombotic events and noncardiovascular deaths will be identified by the investigative site or through medical review and will be sent to a blinded Clinical Event Committee for adjudication at regular intervals.

#### 9.5. Pharmacokinetics

A venous blood sample will be drawn at the times indicated in the Schedule of Activities (Section 2) (Weeks 0 [first dose, 2 samples], 4, 8, 12, and 16). These blood samples will be used to determine the plasma concentrations of baricitinib using a validated liquid chromatography

tandem mass spectrometry method. Blood samples that will be used for other laboratory assessments (chemistry, hematology, etc.) should be drawn at approximately the same time as the samples drawn to determine plasma concentrations of baricitinib. The timing will be as follows:

- At Visit 2 (Week 0), baseline laboratory samples should be taken before administration of investigational product. Patients will take their investigational product in the clinic, and PK samples will be drawn 15 minutes and 1 hour postdose.
- At Visit 5 (Week 4), patients will be asked to take their investigational product at home prior to visiting the clinic. The clinic visit should be scheduled so that the blood sample collected during this visit is drawn 2 to 4 hours after the dose is taken at home.
- For Visit 6 (Week 8) and Visit 7 (Week 12) patients will be asked to not take their investigational product before visiting the clinic, and a blood sample will be collected at any time predose on the day of the clinic visits. If the patient has taken the oral dose prior to the visit, the sample may be drawn anytime postdose, and the inability to collect a predose sample will not be considered a protocol violation.
- At Visit 8 (Week 16), patients will be asked to take their investigational product at home prior to visiting the clinic. The clinic visit should be scheduled so that the blood sample collected during this visit is drawn 4 to 6 hours after the oral dose is taken at home.
- For the ETV, a sample may be drawn anytime if the last dose of investigational drug was taken within the last 48 hours.

For visits where PK samples will be collected, the actual date and 24-hour clock time of sample collection, and the date and time of the last 2 doses prior to the sample being drawn, should be recorded. At Visit 5 (Week 4) and Visit 8 (Week 16), these 2 doses should be the dose given the morning of the day of sample collection and the dose given the previous day. At Visit 6 (Week 8) and Visit 7 (Week 12), the 2 previous doses should be the dose taken yesterday and the dose taken the day before that.

This sampling schedule should be followed as closely as possible; however, failure to take PK samples at these specified times will not be considered a protocol violation. If the patient fails to follow the directions for a particular visit, the sample should still be collected at that visit, and the date and 24-hour clock time of sample collection and the date and time of the 2 doses prior to the sample being drawn should be recorded.

Only samples from patients receiving baricitinib will be assayed; samples from patients receiving placebo will not be assayed. Pharmacokinetic samples will be kept in storage at a laboratory facility designated by the sponsor. Pharmacokinetic samples may also be assayed for additional exploratory analyses. Pharmacokinetic results will not be provided to investigative sites until the completion of the study or to the blinded study team until the study has been unblinded.

Bioanalytical samples collected to measure investigational product concentration will be retained for a maximum of 1 year following last patient visit for the study.

## 9.6. Pharmacodynamics

Not applicable.

## 9.7. Pharmacogenetics

## 9.7.1. Blood Samples for Pharmacogenetic Research

A blood sample will be collected for pharmacogenetic analysis as specified in the Schedule of Activities (Section 2) where local regulations allow.

There is growing evidence that genetic variation may impact a patient's response to therapy. Variable response to therapy may be due to genetic determinants that impact drug absorption, distribution, metabolism, and excretion, the mechanism of action of the drug, the disease etiology, and/or the molecular subtype of the disease being treated. In the event of an unexpected AE, the samples may be genotyped and analysis may be performed to evaluate a genetic association with response to baricitinib. These investigations may be limited to targeted exome sequencing approach of known targets involved in drug metabolism or, if appropriate, genome-wide association studies may be performed to identify regions of the genome associated with the variability observed in drug response. Samples will only be used for investigations related to disease and drug or class of drugs under study in the context of this clinical program.

Samples will not be used to conduct unspecified disease or population genetic research either now or in the future. Samples will be used to investigate variable response to baricitinib and to investigate genetic variants thought to play a role in AD or other inflammatory skin diseases. Assessment of variable response may include evaluation of AEs or differences in efficacy.

All samples will be coded with the patient number. These samples and any data generated can be linked back to the patient only by the investigator site personnel.

Samples will be retained for a maximum of 15 years after the last patient visit for the study, or for a shorter period if local regulations and/or (ethical review boards (ERBs)/investigational review boards) impose shorter time limits, at a facility selected by Lilly. This retention period enables use of new technologies, response to regulatory questions, and investigation of variable response that may not be observed until later in the development of baricitinib or after baricitinib becomes commercially available.

Molecular technologies are expected to improve during the 15-year storage period and therefore cannot be specifically named. However, existing approaches include whole genome or exome sequencing, genome-wide association studies, and candidate gene studies. Regardless of technology utilized, genotyping data generated will be used only for the specific research scope described in this section.

#### 9.8. Biomarkers

Biomarker research is performed to address questions of relevance to drug disposition, target engagement, pharmacodynamics (PD), mechanism of action, variability of patient response (including safety), and clinical outcome. Sample collection is incorporated into clinical studies to enable examination of these questions through measurement of biomolecules including DNA, RNA, proteins, lipids, and other cellular elements.

Blood samples for nonpharmacogenetic biomarker research will be collected at the times specified in the Schedule of Activities (Section 2) where local regulations allow.

Samples will be used for research on the drug target, disease process, variable response to baricitinib, pathways associated with AD, mechanism of action of baricitinib, and/or research method or in validating diagnostic tools or assay(s) related to AD.

All samples will be coded with the patient number. These samples and any data generated can be linked back to the patient only by the investigator site personnel.

Samples will be retained for a maximum of 15 years after the last patient visit for the study, or for a shorter period if local regulations and ERBs impose shorter time limits, at a facility selected by Lilly. This retention period enables use of new technologies, response to regulatory questions, and investigation of variable response that may not be observed until later in the development of baricitinib or after baricitinib becomes commercially available.

### 9.9. Medical Resource Utilization and Health Economics

Health Economics will be evaluated in this study utilizing the EQ-5D-5L and WPAI-AD (see Section 9.1.3). Medical Resource Utilization parameters will not be evaluated in this study.

## 10. Statistical Considerations

## 10.1. Sample Size Determination

Study JAHL will aim to enroll approximately 600 patients ≥18 years of age. The proposed sample size will ensure a >90% power to detect an absolute difference of 20% between the baricitinib 4-mg and placebo treatment groups and the baricitinib 2-mg and placebo treatment groups, each using a 2-sided alpha of 0.025, assuming a 10% placebo response rate for the primary endpoint. The assumptions are based on what was observed in the Phase 2 study (JAHG). The proposed end point of IGA 0 or 1 represents patients whose AD is clear or almost clear from a baseline of moderate or severe disease. The anticipated effect size represents 3 times more patients achieving this benefit compared to placebo, which, in discussion with therapeutic experts, is of a magnitude that is considered clinically relevant.

Sample size and power estimates were obtained from nQuery® Advisor 7.0.

## 10.2. Populations for Analyses

Unless otherwise specified, the efficacy and health outcome analyses will be conducted on the intent-to-treat population, defined as all randomized patients, even if the patient does not receive the correct treatment, or otherwise did not follow the protocol. Patients will be analyzed according to the treatment to which they were assigned. Significant protocol violations will be described in the SAP.

Safety analyses will be done on all randomized patients who receive at least 1 dose of investigational product and who did not discontinue from the study for the reason "Lost to Follow-up" at the first postbaseline visit.

Further details of other populations will be described in the SAP. Patients will be analyzed according to the dosing regimen to which they were assigned in the Treatment Period.

# 10.3. Statistical Analyses

#### 10.3.1. General Statistical Considerations

Statistical analysis of this study will be the responsibility of Lilly or its designee. A detailed SAP describing the statistical methodologies will be developed by Lilly or its designee.

Any change to the data analysis methods described in the protocol will require an amendment ONLY if it changes a principal feature of the protocol. Any other change to the data analysis methods described in the protocol, and the justification for making the change, will be described in the clinical study report (CSR). Additional exploratory analyses of the data will be conducted as deemed appropriate.

All tests of treatment effects will be conducted at a 2-sided alpha level of 0.05, unless otherwise stated. Treatment comparisons of discrete efficacy variables between baricitinib and placebo will be made using a logistic regression analysis with region, disease severity, and treatment group in the model. The percentages, difference in percentages, and 95% confidence interval

(CI) of the difference in percentages will be reported. Treatment-by-region interaction will be added to the logistic regression model of the primary and key secondary variables as a sensitivity analysis. If this interaction is significant at a 2-sided 0.1 level, further inspection will be used to assess whether the interaction is quantitative (i.e., the treatment effect is consistent in direction but not size of effect) or qualitative (the treatment is beneficial for some but not all regions). The p-value from the Fisher exact test will also be produced.

When evaluating continuous measures over time, a restricted maximum likelihood-based mixed-effects model of repeated measures (MMRM) will be used. The model will include treatment, region, baseline severity, visit, and treatment-by-visit interaction as fixed categorical effects and baseline score and baseline score-by-visit interaction as fixed continuous effects. An unstructured (co)variance structure will be used to model the between- and within-patient errors. If this analysis fails to converge, other structures will be tested. The Kenward–Roger method will be used to estimate the degrees of freedom. Type III sums of squares for the least squares means (LSMs) will be used for the statistical comparison; 95% CI will also be reported. Contrasts will be set up within the model to test treatment groups at specific time points of interest. Further details on the use of MMRM will be described in the SAP.

Treatment comparisons of continuous efficacy and health outcome variables may also be made using analysis of covariance (ANCOVA) with region, disease severity, treatment group, and baseline value in the model. Type III tests for LSM will be used for statistical comparison between treatment groups. The LSM difference, standard error, p-value, and 95% CI may also be reported. The method used to handle missing data will be specified in the SAP.

Fisher exact test will be used for the AEs, discontinuation, and other categorical safety data for between-treatment group comparisons. Continuous vital signs, body weight, and other continuous safety variables including laboratory variables will be analyzed by an ANCOVA with treatment and baseline value in the model. Shift tables for categorical safety analyses (e.g., "high" or "low" laboratory results) will also be produced.

#### Missing data imputation:

- 1. Nonresponder imputation (NRI): All patients who discontinue the study or the study treatment at any time for any reason will be defined as nonresponders for the NRI analysis for categorical variables such as IGA 0/1 or EASI 50/75/90 after discontinuation and onward. Patients who receive rescue therapy will be analyzed as nonresponders after rescue and onward. An additional analysis will be performed that includes all available data whether rescue medication was given or not.
- 2. MMRM: Continuous variables such as EASI and SCORAD scores will be assumed to be missing after rescue or discontinuation and then an MMRM analysis will be performed. An additional analysis will be performed that includes all available data whether rescue medication was given or not.
- 3. Last observed carried forward (LOCF): An additional analysis will be performed that uses the last observed value on or prior to discontinuation or rescue therapy. This will

then be analyzed using a logistic model for categorical variables or ANCOVA for continuous variables as described above.

Additional sensitivity analyses for the primary and key secondary endpoints such as tipping point analyses as well as a reference based multiple imputation method may be done and will be specified in the SAP.

#### **Adjustment for Multiple Comparisons:**

Multiplicity controlled analyses will be performed on the primary and major secondary endpoints to control the overall family-wise Type I error rate at a 2-sided  $\alpha$  level of 0.05. The graphical multiple testing procedure described in Bretz et al. (2011) will be used. The graphical approach is a closed testing procedure; hence it strongly controls the family-wise error rate across all endpoints (Alosh et al. 2014). Details of the specific graphical testing scheme (including testing order, interrelationships, Type I error allocation, and the associated propagation) will be prespecified in the SAP.

The following is a list of primary and key secondary endpoints to be tested:

#### Primary:

- proportion of baricitinib 4-mg patients achieving IGA of 0 or 1 and ≥2-point improvement from baseline at Week 16.
- proportion of baricitinib 2-mg patients achieving IGA of 0 or 1 and ≥2-point improvement from baseline at Week 16.

#### **Key Secondaries:**

• proportion of baricitinib 1-mg patients achieving IGA of 0 or 1 with a  $\geq$ 2-point improvement at Week 16.

Evaluated for 1-mg, 2-mg, and 4-mg:

- proportion of patients achieving EASI75 at 16 weeks
- proportion of patients achieving EASI90 at 16 weeks
- percent change from baseline in EASI score at 16 weeks
- proportion of patients achieving SCORAD75 at 16 weeks
- proportions of patients achieving a 4-point improvement in Itch NRS at 1 week, 2 weeks, 4 weeks, and 16 weeks
- mean change from baseline in the score of Item 2 from the ADSS at 1 week and 16 weeks
- mean change from baseline in skin pain NRS at 16 weeks.

## 10.3.2. Treatment Group Comparability

## 10.3.2.1. Patient Disposition

All patients who discontinue from the study or the study treatment will be identified, along with their reason for discontinuation. Reasons for discontinuation from the study will be summarized by treatment group.

#### 10.3.2.2. Patient Characteristics

Demographic and baseline characteristics will be summarized descriptively by treatment group. Descriptive statistics including number of patients, mean, standard deviation, median, minimum, and maximum will be provided for continuous measures, and frequency counts and percentages will be tabulated for categorical measures. No formal statistical comparisons will be made among treatment groups unless otherwise stated.

#### 10.3.2.3. Concomitant Therapy

Concomitant medications will be descriptively summarized by treatment group in terms of frequencies and percentages using the safety population. The medications will be coded accordingly.

### 10.3.2.4. Treatment Compliance

Treatment compliance with the randomly assigned study medication will be evaluated at every clinic visit through the counts of returned investigational product tablets. A patient will be considered significantly noncompliant if he or she misses more than 20% of the prescribed doses during the study, unless the patient's investigational product is withheld by the investigator for safety reasons; that is, compliance <80%. Similarly, a patient will be considered significantly noncompliant if he or she is judged by the investigator to have intentionally or repeatedly taken more than the prescribed amount of medication, that is, compliance  $\ge 120\%$ .

# 10.3.3. Efficacy Analyses

## 10.3.3.1. Primary Analyses

The primary efficacy measure is the binary outcome of response defined as IGA score of 0 or 1 (clear or almost clear skin) and ≥2-point improvement from baseline at Week 16. Primary analysis will be conducted using a logistic regression as described above with treatment and the stratification variables (disease severity and region) in the model. Nonresponder imputation for missing data as described above will be used.

Additional analysis of the primary efficacy outcome will include analyzing the outcome as observed, that is, whether or not rescue medication was used.

## 10.3.3.2. Secondary Analyses

The following secondary categorical outcomes will be analyzed in a similar manner as the primary, that is, using the same logistic regression model. Nonresponder imputation will be used for these analyses unless otherwise noted.

- EASI75 at Week 16. EASI75 is defined as having an improvement of at least 75% from baseline. Besides NRI, this outcome will also be analyzed using observed cases, that is, whether rescue medication was given or not.
- EASI90 at Week 16. EASI90 is defined as having an improvement of at least 90% from baseline.
- SCORAD75 at Week 16. SCORAD75 is defined as having an improvement of at least 75% from baseline
- SCORAD90 at Week 16. SCORAD90 is defined as having an improvement of at least 90% from baseline.
- 4-point improvement in Itch NRS at 1 week, 2 weeks, 4 weeks, and 16 weeks.

The following continuous measures will be analyzed with the MMRM model described above unless otherwise noted. Contrasts within the MMRM model will be used to assess treatment differences for time points of interest as specified above in the list of objectives.

- Mean change from baseline in the following outcome measures:
  - o ADSS Item 2 score
  - EASI score
  - SCORAD score
  - o BSA
  - o Itch NRS
  - POEM total score
  - o PGI-S-AD
  - o HADS
  - o DLOI total score
  - o WPAI
  - o EQ-5D-5L.

The EASI total score and SCORAD total score will also be analyzed as observed, that is, not assuming missing values after rescue medication is given.

# 10.3.4. Safety Analyses

All safety data will be descriptively summarized by treatment groups and analyzed using the safety population.

Treatment-emergent adverse events (TEAEs) are defined as AEs that first occurred or worsened in severity after the first dose of study treatment. The number of TEAEs as well as the number and percentage of patients who experienced at least 1 TEAE will be summarized using MedDRA (Medical Dictionary for Regulatory Activities) for each system organ class (or a body system) and each preferred term by treatment group. Serious adverse events and AEs that lead to discontinuation of investigational product will also be summarized by treatment group. Fisher exact test will be used to perform comparisons between each baricitinib dose and the placebo group.

All clinical laboratory results will be descriptively summarized by treatment group. Individual results that are outside of normal reference ranges will be flagged in data listings. Quantitative clinical hematology, chemistry, and urinalysis variables obtained at the baseline to postbaseline visits will be summarized as changes from baseline by treatment group and analyzed using ANCOVA with treatment and baseline value in the model. Categorical variables, including the incidence of abnormal values and incidence of adverse events of special interest, will be summarized by frequency and percentage of patients in corresponding categories. Shift tables will be presented for selected measures.

Observed values and changes from baseline (predose or screening if missing) for vital signs and physical characteristics will be descriptively summarized by treatment group and time point. Change from baseline to postbaseline in vital signs and body weight will be analyzed using ANCOVA with treatment and baseline value in the model.

The incidence and average duration of investigational product interruptions will be summarized and compared descriptively among treatment groups. Various techniques may be used to estimate the effects of investigational product interruptions on safety measures. Further analyses may be performed and will be planned in the SAP.

Data collected after initiation of rescue therapy will be summarized as appropriate.

## 10.3.5. Pharmacokinetic/Pharmacodynamic Analyses

All plasma baricitinib concentration—time data will be pooled and evaluated using population PK methods. A covariate screen of patient and study-specific factors will be included in the analyses based on factors investigated in previous and (if any) ongoing PK analyses, and on their relevance to the target population. Exploratory and/or model-based analyses examining the relationships between baricitinib exposure and efficacy and response endpoints will be conducted. Other analyses of efficacy and safety outcome measures may also be assessed as scientifically appropriate and warranted by available data. Details about the analyses to be conducted will be contained in the PK/PD analysis plan.

# 10.3.6. Other Analyses

#### 10.3.6.1. Health Outcome Measures

The health outcome measures will be analyzed using methods described for continuous or categorical data as described for efficacy measures in Section 10.3.3.

## 10.3.6.2. Subgroup Analyses

To assess whether the treatment effect is similar across subgroups for the primary efficacy outcome, a logistic model will be used and will include treatment, stratification variables, the subgroup variable (e.g., sex) and the subgroup by treatment interaction. If the interaction is statistically significant at  $\alpha$ =0.10, the nature of the interaction will be explored, that is, within each subgroup the treatment effect will be estimated. Similarly, for the continuous variables of EASI, the MMRM model will include additional variables for subgroup and the subgroup by treatment interaction.

Subgroups to be evaluated will include region, baseline severity, sex, age, race, prior therapy, etc. Further definitions for the levels of the subgroup variables, the analysis methodology, and any additional subgroup analyses will be defined in the SAP. Because this study is not powered for subgroup analyses, all subgroup analyses will be treated as exploratory.

## 10.3.7. Interim Analyses

#### 10.3.7.1. Data Monitoring Committee

A DMC will oversee the conduct of this trial. The DMC will consist of members external to Lilly. This DMC will follow the rules defined in the DMC charter, focusing on potential and identified risks for this molecule and for this class of compounds. Data Monitoring Committee membership will include, at a minimum, specialists with expertise in dermatology, statistics, and other appropriate specialties.

The DMC will be authorized to review unblinded results of analyses by treatment group prior to database lock, including study discontinuation data, AEs including SAEs, clinical laboratory data, vital sign data, etc. The DMC may recommend continuation of the study, as designed; temporary suspension of enrollment; or the discontinuation of a particular dose regimen or the entire study. While the DMC may request to review efficacy data to investigate the benefit/risk relationship in the context of safety observations for ongoing patients in the study, no information regarding efficacy will be communicated. Moreover, the study will not be stopped for positive efficacy results nor will it be stopped for futility. Hence, no alpha is spent. Details of the DMC, including its operating characteristics, will be documented in a DMC charter and DMC analysis plan.

Besides DMC members, a limited number of pre-identified individuals may gain access to the limited unblinded data, as specified in the unblinding plan, prior to the interim or final database lock to initiate the final population PK/PD model development processes or for preparation of regulatory documents. Information that may unblind the study during the analyses will not be reported to study sites or blinded study team until the study has been unblinded.

Unblinding details will be specified in a separate unblinding plan document.

#### 10.3.7.2. Adjudication Committee

A blinded Clinical Event Committee will adjudicate potential MACE (cardiovascular death, MI, stroke), other cardiovascular events (such as hospitalization for unstable angina, hospitalization for heart failure, serious arrhythmia, resuscitated sudden death, cardiogenic shock, coronary revascularization such as coronary artery bypass graft or percutaneous coronary intervention), venous thrombotic events, and noncardiovascular deaths. Details of membership, operations, recommendations from the Committee, and the communication plan will be documented in the Charter.

## 11. References

- Alosh M, Bretz F, Huque M. Advanced multiplicity adjustment methods in clinical trials. *Stat Med.* 2014;33(4):693-713.
- Basra MK, Salek MS, Camilleri L, Sturkey R, Finlay AY. Determining the minimal clinically important difference and responsiveness of the Dermatology Life Quality Index (DLQI): further data. *Dermatology*. 2015;230(1):27-33.
- Bieber, T. Atopic Dermatitis. *Ann Derm.* 2010;22(2):125-137.
- Bieber T, Straeter B. Off-label prescriptions for atopic dermatitis in Europe. *Allergy*. 2015;70(1):6-11.
- Bretz F, Posch M, Glimm E, Klinglmueller F, Maurer W, Rohmeyer K. Graphical approaches for multiple comparison procedures using weighted Bonferroni, Simes, or parametric tests. *Biom J.* 2011;53(6):894-913.
- Charman CR, Venn AJ, Williams, HC. The Patient-Oriented Eczema Measure. *Arch Dermatol.* 2004:140:1513-1519.
- Clark JD, Flanagan ME, Telliez JB. Discovery and development of Janus kinase (JAK) inhibitors for inflammatory diseases. *J Med Chem.* 2014;57(12):5023-5038.
- Divekar R, Kita H. Recent advances in epithelium-derived cytokines (IL-33, IL-25, and thymic stromal lymphopoietin) and allergic inflammation. *Curr Opin Allergy Clin Immunol*. 2015;15(1):98-103.
- Dougados M, van der Heijde D, Chen YC, Greenwald M, Drescher E, Liu J, Beattie S, Witt S, de la Torre I, Gaich C, Rooney T, Schlichting D, de Bono S, Emery P. Baricitinib in patients with inadequate response or intolerance to conventional synthetic DMARDs: results from the RABUILD study. *Ann Rheum Dis.* 2017;76(1):88-95.
- Eichenfield LF, Tom WL, Chamlin SL, Feldman SR, Hanifin JM, Simpson EL, Berger TG, Bergman JN, Cohen DE, Cooper KD, Cordoro KM, Davis DM, Krol A, Margolis DJ, Paller AS, Schwarzenberger K, Silverman RA, Williams HC, Elmets CA, Block J, Harrod CG, Smith Begolka W, Sidbury R. Guidelines of care for the management of atopic dermatitis: section 1. Diagnosis and assessment of atopic dermatitis. *J Am Acad Dermatol*. 2014;70(2):338-3351.
- EuroQol Group. EQ-5D-5L User Guide. Version 2.1. Available at: http://www.euroqol.org/fileadmin/user\_upload/Documenten/PDF/Folders\_Flyers/EQ-5D-5L UserGuide 2015.pdf. April 2015. Accessed March 2017.
- Fleischmann R, Schiff M, van der Heijde D, Ramos-Remus C, Spindler A, Stanislav M, Zerbini CA, Gurbuz S, Dickson C, de Bono S, Schlichting D, Beattie S, Kuo WL, Rooney T, Macias W, Takeuchi T. Baricitinib, methotrexate, or combination in patients with rheumatoid arthritis and no or limited prior disease-modifying antirheumatic drug treatment. *Arthritis Rheumatol*. 2017;69(3):506-517.
- Fridman JS, Scherle PA, Collins R, Burn TC, Li Y, Li J, Covington MB, Thomas B, Collier P, Favata MF, Wen X, Shi J, McGee R, Haley PJ, Shepard S, Rodgers JD, Yeleswaram S, Hollis G, Newton RC, Metcalf B, Friedman SM, Vaddi K. Selective inhibition of JAK1 and JAK2 is

- efficacious in rodent models of arthritis: preclinical characterization of INCB028050. *J Immunol*. 2010;184(9):5298-5307.
- Futamura M, Leshem YA, Thomas KS, Nankervis H, Williams HC, Simpson EL. A systematic review of Investigator Global Assessment (IGA) in atopic dermatitis (AD) trials: Many options, no standards. *J Am Acad Dermatol*. 2016;74(2):288-294.
- Genovese MC, Kremer J, Zamani O, Ludivico C, Krogulec M, Xie L, Beattie SD, Koch AE, Cardillo TE, Rooney TP, Macias WL, de Bono S, Schlichting DE, Smolen JS. Baricitinib in patients with refractory rheumatoid arthritis. *N Engl J Med*. 2016;374(13):1243-1252.
- Hanifin JM, Thurston M, Omoto M, Cherill R, Tofte SJ, Graeber M. The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. EASI Evaluator Group. *Exp Dermatol.* 2001;10(1):11-18.
- Herdman M, Gudex C, Lloyd A, Janssen MF, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). *Qual Life Res.* 2011;20(10):1727-1736.
- Hongbo Y, Thomas CL, Harrison MA, Salek MS, Finlay AY. Translating the science of quality of life into practice: What do dermatology life quality index scores mean? *J Invest Dermatol*. 2005;125(4):659-664.
- Khilji FA, Gonzalez M, Finlay AY. Clinical meaning of change in Dermatology Life Quality Index scores. *Br J Dermatol*. 2002;147(suppl 62):25-54.
- Kimball AB, Naegeli AN, Edson-Heredia E, Lin CY, Gaich C, Nikai E, Yosipovitch G. Psychometric properties of the Itch Numeric Rating Scale in patients with moderate-to-severe plaque psoriasis. *Br J Dermatol.* 2016;175(1):157-162.
- Krakowski AC, Eichenfield LF, Dohil MA. Management of atopic dermatitis in the pediatric population. *Pediatrics*. 2008;122(4):812-824.
- Kunz B, Oranje AP, Labrèze L, Stadler JF, Ring J, Taïeb A. Clinical validation and guidelines for the SCORAD index: consensus report of the European Task Force on Atopic Dermatitis. *Dermatology*. 1997;195(1):10-19.
- Langenbruch A, Radtke M, Franzke N, Ring J, Foelster-Holst R, Augustin M. Quality of health care of atopic eczema in Germany: results of the national health care study AtopicHealth. *J Eur Acad Dermatol Venereol*. 2014;28(6):719-726.
- Langley RG, Feldman SR, Nyirady J, van de Kerkhof P, Papavassilis C. The 5-point Investigator's Global Assessment (IGA) Scale: A modified tool for evaluating plaque psoriasis severity in clinical trials. *J Dermatolog Treat*. 2015;26(1):23-31.
- Li M, Messaddeq N, Teletin M, Pasquali JL, Metzger D, Chambon P. Retinoid X receptor ablation in adult mouse keratinocytes generates an atopic dermatitis triggered by thymic stromal lymphopoietin. *Proc Natl Acad Sci U S A*. 2005;102(41):14795-14800.
- Mallinckrodt CH, Tamura RN, Tanaka Y. Recent developments in improving signal detection and reducing placebo response in psychiatric clinical trials. *J Psychiatric Res*. 2011;45:1202-1207

- Moniaga CS, Jeong SK, Egawa G, Nakajima S, Hara-Chikuma M, Jeon JE, Lee SH, Hibino T, Miyachi Y, Kabashima K. Protease activity enhances production of thymic stromal lymphopoietin and basophil accumulation in flaky tail mice. *Am J Pathol*. 2013;182(3):841-851.
- Naegeli AN, Flood E, Tucker J, Devlen J, Edson-Heredia E. The Worst Itch Numeric Rating Scale for patients with moderate to severe plaque psoriasis or psoriatic arthritis. *Int J Dermatol.* 2015;54(6):715-722.
- Nomura T, Kabashima K. Advances in atopic dermatitis in 2015. *J Allergy Clin Immunol*. 2015;138(6):1548-1555.
- Palmer CN, Irvine AD, Terron-Kwiatkowski A, Zhao Y, Liao H, Lee SP, Goudie DR, Sandilands A, Campbell LE, Smith FJ, O'Regan GM, Watson RM, Cecil JE, Bale SJ, Compton JG, DiGiovanna JJ, Fleckman P, Lewis-Jones S, Arseculeratne G, Sergeant A, Munro CS, El Houate B, McElreavey K, Halkjaer LB, Bisgaard H, Mukhopadhyay S, McLean WH. Common loss-of-function variants of the epidermal barrier protein filaggrin are a major predisposing factor for atopic dermatitis. *Nat Genet.* 2006;38:441-446.
- Papp KA, Menter MA, Raman M, Disch D, Schlichting DE, Gaich C, Macias W, Zhang X, Janes JM. A randomized phase 2b trial of baricitinib, an oral Janus kinase (JAK) 1/JAK2 inhibitor, in patients with moderate-to-severe psoriasis. *Br J Dermatol*. 2016;174(6):1266-1276.
- Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. *Pharmacoeconomics*. 1993;4(5):353-365.
- Schram ME, Spuls PI, Leeflang MM, Lindeboom R, Bos JD, Schmitt J. EASI, (objective) SCORAD and POEM for atopic eczema: responsiveness and minimal clinically important difference. *Allergy*. 2012;67(1):99-106. Epub 2011 Sep 27.
- Simpson EL. Comorbidity in atopic dermatitis. Curr Dermatol Rep. 2012;1(1):29-38.
- Snaith RP. The Hospital Anxiety and Depression Scale. *Health and Quality of Life Outcomes*. 2003;1:29. Available at: http://www.hqlo.com/content/1/1/29. Accessed February 2017.
- Stalder JF, Taïeb A, Atherton DJ, et al. for the European Task Force on Atopic Dermatitis. Severity scoring of atopic dermatitis: the SCORAD index. Consensus Report of the European Task Force on Atopic Dermatitis. *Dermatology*. 1993;186(1):23-31.
- Tadicherla S, Ross K, Shenefelt PD, Fenske NA. Topical Corticosteroids in Dermatology. *J Drugs Dermatol.append* 2009;8(12):1093-1105.
- Taylor PC, Keystone EC, van der Heijde D, Weinblatt ME, del Carmen Morales L, Gonzaga JR, Yakushin S, Ishii T, Emoto K, Beattie S, Arora V, Gaich CL, Rooney T, Schlichting D, Macias WL, de Bono S, Tanaka. Baricitinib versus placebo or adalimumab in rheumatoid arthritis. *N Engl J Med.* 2017;376:652-662.
- Tuttle KR, Brosius FC, Adler SG, Kretzler M, Mehta RL, Tumlin JA, Liu J, Silk ME, Cardillo TE, Duffin KL, Haas JV, Macias WL, Janes JM. Baricitinib in diabetic kidney disease: Results from a Phase 2, multicenter, randomized, double-blind, placebo-controlled study. Paper presented at: Annual Meeting of the American Diabetes Association; 5–9 June 2015; Boston, MA.

- Vaddi K, Luchi M. JAK inhibition for the treatment of rheumatoid arthritis: a new era in oral DMARD therapy. *Expert Opin Investig Drugs*. 2012;21(7):961-973.
- White D, Leach C, Sims R, Atkinson M, Cottrell D. Validation of the Hospital Anxiety and Depression Scale for use with adolescents. *Br J Psychiatry*. 1999;175(5):452-454.
- [WHO] World Health Organization. Model Prescribing Information: Drugs used in skin diseases. 1997; Geneva.
- Wilson SR, Thé L, Batia LM, Beattie K, Katibah GE, McClain SP, Pellegrino M, Estandian DM, Bautista DM. The epithelial cell-derived atopic dermatitis cytokine TSLP activates neurons to induce itch. *Cell*. 2013;155(2):285-295.
- Yano C, Saeki H, Ishiji T, Ishiuji Y, Sato J, Tofuku Y, Nakagawa H. Impact of disease severity on sleep quality in Japanese patients with atopic dermatitis. *J Dermatol Sci*. 2013;72(2):195-197.
- Ziegler SF, Roan F, Bell BD, Stoklasek TA, Kitajima M, Han H. The biology of thymic stromal lymphopoietin (TSLP). *Adv Pharmacol*. 2013;66:129-155.
- Zigmond AS, Snaith RP. The Hospital Anxiety and Depression Scale. *Acta Psychiatr Scand*. 1983;67:361-370.
## 12. Appendices

## **Appendix 1. Abbreviations and Definitions**

| Term | Definition |
|---|---|
| AD | atopic dermatitis |
| ADSS | Atopic Dermatitis Sleep Scale |
| AE | adverse event: Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. |
| ALT | alanine aminotransferase |
| ALP | alkaline phosphatase |
| ANCOVA | analysis of covariance |
| AST | aspartate aminotransferase |
| blinding/masking | A single-blind study is one in which the investigator and/or his staff are aware of the treatment but the patient is not, or vice versa, or when the sponsor is aware of the treatment but the investigator and/his staff and the patient are not. A double-blind study is one in which neither the patient nor any of the investigator or sponsor staff who are involved in the treatment or clinical evaluation of the subjects are aware of the treatment received. |
| BSA | body surface area |
| СІ | confidence interval |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CSR | clinical study report |
| DLQI | Dermatology Life Quality Index |
| DMC | data monitoring committee |
| DNA | deoxyribonucleic acid |
| DVT | deep vein thrombosis |
| EASI | Eczema Area and Severity Index |
| ECG | electrocardiogram |

eCOA electronic clinical outcome assessment

**eCRF** electronic case report form

**eGFR** estimated glomerular filtration rate

enroll The act of assigning a patient to a treatment. Patients who are enrolled in the trial are

those who have been assigned to a treatment.

**Enter** Patients entered into a trial are those who sign the informed consent form directly or

through their legally acceptable representatives.

EQ-5D-5L European Quality of Life-5 Dimensions-5 Levels

**ERB** ethical review board

**ETV** early termination visit

**FDA** the Food and Drug Administration

**GCP** good clinical practice

**HADS** Hospital Anxiety Depression Scale

**HBsAg** hepatitis B surface antigen

**HBV** hepatitis B virus

**HCV** hepatitis C virus

HIV human immunodeficiency virus

ΙB Investigator's Brochure

**ICF** informed consent form

ICH International Council for Harmonisation

**IGA** Investigator's Global Assessment

IL interleukin

interim analysis An interim analysis is an analysis of clinical study data, separated into treatment groups,

that is conducted before the final reporting database is created/locked.

**INR** international normalized ratio

Investigational

A pharmaceutical form of an active ingredient or placebo being tested or used as a product reference in a clinical trial, including products already on the market when used or

assembled (formulated or packaged) in a way different from the authorized form, or marketed products used for an unauthorized indication, or marketed products used to

gain further information about the authorized form.

**IWRS** interactive web-response system **JAK** Janus kinase

**LOCF** last observed carried forward

**LSM** least squares mean

**MACE** major adverse cardiovascular events

MI myocardial infarction

**MMRM** mixed-effects model of repeated measures

**NRI** nonresponder imputation

NRS Numeric Rating Scale

PD pharmacodynamics(s)

**PDE-4 inhibitor** phosphodiesterase type 4 inhibitor

**PK** pharmacokinetic(s)

POEM Patient-Oriented Eczema Measure

**PPD** purified protein derivative

**PRO/ePRO** patient-reported outcomes/electronic patient-reported outcomes

**QD** once daily

**QoL** quality of life

**SAE** serious adverse event

**SAP** statistical analysis plan

SCORAD SCORing Atopic Dermatitis

**STAT** signal transducer and activator of transcription

**SUSAR** suspected unexpected serious adverse reaction

TB tuberculosis

**TBL** total bilirubin level

TCNI topical calcineurin inhibitor

TCS topical corticosteroids

**TEAE** Treatment-emergent adverse event: An untoward medical occurrence that emerges

during a defined treatment period, having been absent pretreatment, or worsens relative to the pretreatment state, which does not necessarily have to have a causal relationship

with this treatment.

**TSH** thyroid-stimulating hormone

**TSLP** thymic stromal lymphopoietin

VAS Visual Analog Scale

vlGA-AD validated Investigator's Global Assessment for Atopic Dermatitis

**VTE** venous thromboembolic event (deep vein thrombosis or pulmonary embolism)

**WPAI-AD** The Work Productivity and Activity Impairment–Atopic Dermatitis

#### **Appendix 2. Clinical Laboratory Tests**

Hematology<sup>a,b</sup> Clinical Chemistry<sup>a,b</sup>
Hemoglobin Serum Concentrations of:

Hematocrit Sodium

Erythrocyte count (RBC) Potassium

Absolute Reticulocyte Count Total bilirubin

Mean cell volume Direct bilirubin

Mean cell hemoglobin Alkaline phosphatase

Mean cell hemoglobin concentration

Leukocytes (WBC)

Alanine aminotransferase (ALT)

Aspartate aminotransferase (AST)

Blood urea nitrogen (BUN)

Absolute counts of:CreatinineNeutrophils, segmentedCystatin CNeutrophils, juvenile (bands)Uric acidLymphocytesCalciumMonocytesGlucoseEosinophilsAlbuminBasophilsTotal protein

Estimated glomerular filtration rate (eGFR)e

Urinalysis<sup>a,b,d</sup> Creatine phosphokinase (CPK)

Color

Specific gravity Other Tests<sup>a</sup>

pH Hepatitis B Surface antigen (HBsAg)<sup>f</sup>
Protein Anti-Hepatitis B Core antibody (HBcAb)<sup>f</sup>

Glucose HBV DNAk

Ketones Anti-Hepatitis B Surface antibody (HBsAb)<sup>f</sup>
Bilirubin Human immunodeficiency virus (HIV)<sup>f</sup>

Urobilinogen Hepatitis C antibody<sup>f</sup>,g

Blood Thyroid-stimulating hormone (TSH)

Leukocyte esterase Exploratory storage samples (serum, plasma and mRNA)

Nitrite Pregnancy Testh

Follicle-stimulating hormonef,i

Lipidsa,cSerum immunoglobulin (IgA, IgG, IgM, and IgE)Total cholesterolQuantiFERON®-TB Gold or T-SPOT®.TB j

Low-density lipoprotein PPD (local testing)
High-density lipoprotein Baricitinib plasma levels

Triglycerides

Abbreviations: FSH = follicle-stimulating hormone; HBV = hepatitis B virus; PPD = purified protein derivative;

RBC = red blood cell; TB = tuberculosis; WBC = white blood cell.

- a Assayed by sponsor-designated laboratory.
- b Unscheduled or repeat blood chemistry, hematology, and urinalysis panels may be performed at the discretion of the investigator, as needed.
- c Fasting lipid profile. Patients should not eat or drink anything except water for 12 hours prior to test. If a patient attends these visits in a nonfasting state, this will not be considered a protocol violation.
- d Microscopic examination of sediment performed only if abnormalities are noted on the routine urinalysis.
- e eGFR for serum creatinine calculated by the central laboratory using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine 2009 equation.
- f Test required at Visit 1 only to determine eligibility of patient for the study.
- g A positive hepatitis C antibody (Hep C antibody) result will be confirmed with an alternate hepatitis C method.
- For all women of childbearing potential, a serum pregnancy test will be performed at Visit 1 and a local urine pregnancy test will be performed at Visit 2 and at all subsequent study visits after Visit 3. If required per local regulations and/or institutional guidelines, pregnancy testing can occur at other times during the study treatment period.
- i To confirm postmenopausal status for women ≥40 and <60 years of age who have had a cessation of menses, an FSH test will be performed. Nonchildbearing potential is defined as an FSH ≥40 mIU/mL and a cessation of menses for at least 12 months.
- J The QuantiFERON®-TB Gold test is the preferred alternative to the PPD test for the evaluation of TB infection, and it may be used instead of the PPD test or T-SPOT®.TB test and may be read locally. If the QuantiFERON® TB Gold test is indeterminate, 1 retest is allowed. If the retest is indeterminate, then the patient is excluded from the study.
- k HBV DNA testing will be done in those patients who are HBcAb+ at screening.

## **Appendix 3. Study Governance Considerations**

# Appendix 3.1. Regulatory and Ethical Considerations, Including the Informed Consent Process

#### Appendix 3.1.1. Informed Consent

The investigator is responsible for ensuring the following:

- that the patient understands the potential risks and benefits of participating in the study.
- that informed consent is given by each patient. This includes obtaining the appropriate signatures and dates on the informed consent form (ICF) prior to the performance of any protocol procedures and prior to the administration of investigational product.
- answering any questions the patient may have throughout the study and sharing in a timely manner any new information that may be relevant to the patient's willingness to continue his or her participation in the trial.

#### Appendix 3.1.2. Ethical Review

The investigator must give assurance that the ERB was properly constituted and convened as required by International Council for Harmonisation (ICH) guidelines and other applicable laws and regulations.

Documentation of ERB approval of the protocol and the ICF must be provided to Lilly before the study may begin at the investigative site(s). Lilly or its representatives must approve the ICF, including any changes made by the ERBs, before it is used at the investigative site(s). All ICFs must be compliant with the ICH guideline on Good Clinical Practice (GCP).

The study site's ERB(s) should be provided with the following:

- the current Investigator Brochure (IB) and updates during the course of the study
- informed consent form
- relevant curricula vitae.

#### Appendix 3.1.3. Regulatory Considerations

This study will be conducted in accordance with:

- consensus ethics principles derived from international ethics guidelines, including the Declaration of Helsinki and Council for International Organizations of Medical Sciences (CIOMS) International Ethical Guidelines
- applicable ICH GCP Guidelines
- applicable laws and regulations.

Some of the obligations of the sponsor will be assigned to a third party.

#### Appendix 3.1.4. Investigator Information

Physicians with a specialty in dermatology will participate as investigators in this clinical trial.

#### Appendix 3.1.5. Protocol Signatures

The sponsor's responsible medical officer will approve the protocol, confirming that, to the best of his or her knowledge, the protocol accurately describes the planned design and conduct of the study.

After reading the protocol, each principal investigator will sign the protocol signature page and send a copy of the signed page to a Lilly representative.

#### Appendix 3.1.6. Final Report Signature

Lilly will select a qualified investigator(s) from among investigators participating in the design, conduct, and/or analysis of the study to serve as the clinical study report (CSR) coordinating investigator. If this investigator is unable to fulfill this function, another investigator will be chosen by Lilly to serve as the CSR coordinating investigator.

The CSR coordinating investigator will sign the final CSR for this study, indicating agreement that, to the best of his or her knowledge, the report accurately describes the conduct and results of the study.

The sponsor's responsible medical officer and statistician will approve the final CSR for this study, confirming that, to the best of his or her knowledge, the report accurately describes the conduct and results of the study.

#### **Appendix 3.2. Data Quality Assurance**

To ensure accurate, complete, and reliable data, Lilly or its representatives will do the following:

- provide instructional material to the study sites, as appropriate
- provide sponsor start-up training to instruct the investigators and study coordinators. This training will give instruction on the protocol, the completion of the CRFs, and study procedures.
- make periodic visits to the study site
- be available for consultation and stay in contact with the study site personnel by mail, telephone, and/or fax
- review and evaluate CRF data and use standard computer edits to detect errors in data collection
- conduct a quality review of the database.

In addition, Lilly or its representatives will periodically check a sample of the patient data recorded against source documents at the study site. The study may be audited by Lilly or its representatives and/or regulatory agencies at any time. Investigators will be given notice before an audit occurs.

The investigator will keep records of all original source data. This might include laboratory tests, medical records, and clinical notes. If requested, the investigator will provide the sponsor, applicable regulatory agencies, and applicable ERBs with direct access to original source documents.

#### Appendix 3.2.1. Data Capture System

An electronic data capture system will be used in this study. The site maintains a separate source for the data entered by the site into the sponsor-provided electronic data capture system.

Electronic patient-reported outcome (ePRO) measures (e.g., a rating scale) and Electronic clinical outcome assessments (eCOAs) are entered into an ePRO/eCOA instrument at the time that the information is obtained. In these instances where there is no prior written or electronic source data at the site, the ePRO/eCOA instrument record will serve as the source.

If ePRO/eCOA records are stored at a third-party site, investigator sites will have continuous access to the source documents during the study and will receive an archival copy at the end of the study for retention.

Any data for which the ePRO/eCOA instrument record will serve to collect source data will be identified and documented by each site in that site's study file.

Case report form data will be encoded and stored in InForm. Data managed by a central vendor, such as laboratory test data, will be stored electronically in the central vendor's database system. Data will subsequently be transferred from the central vendor to the Lilly data warehouse.

Data managed by a central vendor, such as laboratory test data, will be stored electronically in the central vendor's database system. Data will subsequently be transferred from the central vendor to the Lilly data warehouse.

Data from complaint forms submitted to Lilly will be encoded and stored in the global product complaint management system.

#### Appendix 3.3. Study and Site Closure

#### Appendix 3.3.1. Discontinuation of Study Sites

Study site participation may be discontinued if Lilly, the investigator, or the ERB of the study site judges it necessary for medical, safety, regulatory, or other reasons consistent with applicable laws, regulations, and GCP.

#### Appendix 3.3.2. Discontinuation of the Study

The study will be discontinued if Lilly judges it necessary for medical, safety, regulatory, or other reasons consistent with applicable laws, regulations, and GCP.

#### Appendix 4. Hepatic Monitoring Tests For Treatment-Emergent Abnormality

Selected tests may be obtained in the event of a treatment-emergent hepatic abnormality and may be required in follow-up with patients in consultation with the Lilly, its designee, or the clinical research physician.

**Hepatic Monitoring Tests** 

| Hepatic Hematologya | Haptoglobin <sup>a</sup> |
|--------------------------------|--------------------------------------------|
| Hemoglobin | |
| Hematocrit | Hepatic Coagulationa |
| RBC | Prothrombin Time |
| WBC | Prothrombin Time, INR |
| Neutrophils, segmented | |
| Lymphocytes | Hepatic Serologies <sup>a,b</sup> |
| Monocytes | Hepatitis A antibody, total |
| Eosinophils | Hepatitis A antibody, IgM |
| Basophils | Hepatitis B surface antigen |
| Platelets | Hepatitis B surface antibody |
| | Hepatitis B Core antibody |
| Hepatic Chemistry <sup>a</sup> | Hepatitis C antibody |
| Total bilirubin | Hepatitis E antibody, IgG |
| Direct bilirubin | Hepatitis E antibody, IgM |
| Alkaline phosphatase | |
| ALT | Anti-nuclear antibodya |
| AST | |
| GGT | Alkaline Phosphatase Isoenzymesa |
| CPK | - · · · · · |
| | Anti-smooth muscle antibody (or anti-actin |
| | antibody) <sup>a</sup> |

Abbreviations: ALT = alanine aminotransferase; AST = aspirate aminotransferase; CPK = creatinine phosphokinase; GGT = gamma-glutamyl transferase; Ig = immunoglobulin; INR = international normalized ratio; RBC = red blood cell; WBC = white blood cell.

- a Assayed by Lilly-designated or local laboratory.
- b Reflex/confirmation dependent on regulatory requirements and/or testing availability.

# Appendix 5. Liver Function Testing and Hepatic Safety Monitoring

#### **Liver Function Testing and Hepatic Safety Monitoring**

| Analyte | Exclusion<br>Criteria | Additional<br>Hepatic<br>Testing | Hepatic eCRF<br>Reporting | Temporary<br>Interruption of<br>IP | Permanent Discontinuation of IP after Consultation with the Lilly-Designated Medical Monitor |
|---|---|---|---|---|---|
| Protocol<br>Section | Section 6.2 | Section 9.4.9 | Section 9.4.9 | Section 8.1.1 | Section 8.1.2 |
| ALT/AST | ≥2x ULN | ≥3x ULN | ≥5x ULN on ≥2 consecutive tests | ≥5x ULN | <ul> <li>&gt;8x ULN</li> <li>&gt;5x ULN for &gt;2 weeks</li> <li>&gt;3x ULN AND TBL</li> <li>&gt;2x ULN or INR &gt;1.5</li> <li>&gt;3x ULN with</li> <li>symptomsa</li> </ul> |
| ALP | ≥2x ULN | ≥2x ULN | ≥2x ULN on ≥2 consecutive tests | No applicable criteria | <ul> <li>&gt;3x ULN</li> <li>&gt;2.5x ULN AND TBL</li> <li>&gt;2x ULN</li> <li>&gt;2.5x ULN with symptoms<sup>a</sup></li> </ul> |
| TBL | ≥1.5x ULN | ≥2x ULN | ≥2x ULN<br>(excluding<br>Gilbert's<br>syndrome) | No applicable criteria | <ul> <li>ALT &gt;3x ULN AND TBL &gt;2x ULN</li> <li>ALP &gt;2.5x ULN AND TBL &gt;2x ULN</li> </ul> |

Abbreviations: ALP = alkaline phosphatase; ALT = alanine aminotransferase; AST = aspartate aminotransferase; INR = international normalized ratio; IP = investigational product; TBL = total bilirubin level; ULN = upper level of normal.

<sup>&</sup>lt;sup>a</sup> Fatigue, nausea, vomiting, right upper-quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%).

# Appendix 6. American Academy of Dermatology: Criteria for the Diagnosis and Assessment of Atopic Dermatitis

Features to be considered in diagnosis of patients with atopic dermatitis:

#### **Essential Features—Must be present:**

- pruritus
- eczema (acute, subacute, chronic)
  - o typical morphology and age-specific patterns\*
  - o chronic or relapsing history

#### \*Patterns include:

- 1) facial, neck, and extensor involvement in infants and children
- 2)current or previous flexural lesions in any age group
- 3) sparing of the groin and axillary regions

#### Important Features—Seen in most cases, adding support to the diagnosis:

- early age of onset
- atopy
  - o personal and/or family history
  - Immunoglobulin E reactivity
- xerosis

Associated Features—These clinical associations help to suggest the diagnosis of atopic dermatitis but are too nonspecific to be used for defining or detecting atopic dermatitis for research and epidemiologic studies:

- atypical vascular responses (eg, facial pallor, white dermographism, delayed blanch response)
- keratosis pilaris/pityriasis alba/hyperlinear palms/ichthyosis
- ocular/periorbital changes
- other regional findings (e.g., perioral changes/periauricular lesions)
- perifollicular accentuation/lichenification/prurigo lesions

## Exclusionary Features—It should be noted that a diagnosis of atopic dermatitis depends on excluding conditions, such as:

- scabies
- seborrheic dermatitis
- contact dermatitis (irritant or allergic)
- ichthyoses
- cutaneous T-cell lymphoma
- psoriasis
- photosensitivity dermatoses
- immune deficiency diseases
- erythroderma of other causes

Source: Eichenfield et al. Guidelines of care for the management of atopic dermatitis: section 1. Diagnosis and assessment of atopic dermatitis. *J Am Acad Dermatol*. 2014;70(2):338-3351...

# Appendix 7. Classification of Potency for Topical Corticosteroids

| Potency | Potency Class Topical Corticosteroid | | Formulation |
|---|---|---|---|
| Ultra high | I | Clobetasol propionate | Cream 0.05% |
| | | Diflorasone diacetate | Ointment 0.05% |
| High II | | Amcinonide | Ointment 0.1% |
| | | Betamethasone dipropionate | Ointment 0.05% |
| | | Desoximetasone | Cream or ointment 0.025% |
| | | Fluocinonide | Cream, ointment or gel 0.05% |
| | | Halcinonide | Cream 0.1% |
| | III | Betamethasone dipropionate | Cream 0.05% |
| | | Betamethasone valerate | Ointment 0.1% |
| | | Diflorasone diacetate | Cream 0.05% |
| | | Triamcinolone acetonide | Ointment 0.1% |
| Moderate | IV | Desoximetasone | Cream 0.05% |
| | | Fluocinolone acetonide | Ointment 0.025% |
| | | Fludroxycortide | Ointment 0.05% |
| | | Hydrocortisone valerate | Ointment 0.2% |
| | | Triamcinolone acetonide | Cream 0.1% |
| | V | Betamethasone dipropionate | Lotion 0.02% |
| | | Betamethasone valerate | Cream 0.1% |
| | | Fluocinolone acetonide | Cream 0.025% |
| | | Fludroxycortide | Cream 0.05% |
| | | Hydrocortisone butyrate | Cream 0.1% |
| | | Hydrocortisone valerate | Cream 0.2% |
| | | Triamcinolone acetonide | Lotion 0.1% |
| Low | VI | Betamethasone valerate | Lotion 0.05% |
| | | Desonide | Cream 0.05% |
| | | Fluocinolone acetonide | Solution 0.01% |
| | VII | Dexamethasone sodium phosphate | Cream 0.1% |
| | | Hydrocortisone | Lotion, cream, or ointment 2.5% |
| | | Hydrocortisone acetate | Cream 1% |
| | | Methylprednisolone acetate | Cream 0.25% |

Source: WHO (1997) and Tadicherla et al 2009

Appendix 8. Protocol Amendment I4V-MC-JAHL(a)
Summary - A Multicenter, Randomized, Double-Blind,
Placebo-Controlled, Phase 3 Study to Evaluate the
Efficacy and Safety of Baricitinib in Adult Patients with
Moderate to Severe Atopic Dermatitis

#### **Overview**

Protocol I4V-MC-JAHL, A Multicenter, Randomized, Double Blind, Placebo Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Baricitinib in Adult Patients with Moderate to Severe Atopic Dermatitis, has been amended. The new protocol is indicated by amendment (a) and will be used to conduct the study in place of any preceding version of the protocol.

The overall changes and rationale for the changes made to this protocol are described in the following table. Other minor typographical corrections and minor formatting changes not affecting content have been made in the document, and these changes are not identified in the amendment summary table or with strikethrough/underscore.

#### Amendment Summary for Protocol I4V-MC-JAHL Amendment (a)

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| Protocol cover page | Added "BREEZE-AD1" after title of study | Added to associate the alternative study title to the protocol study alias |
| Protocol cover page | Added EudraCT Number | Updated accordingly to align with new protocol template instructions |
| 1. Synopsis | Added IL-4 in discussion section of study rationale | IL-4 also plays a role in the pathogenesis of AD |
| 1. Synopsis | Moved the 2-mg dose from Key Secondary to Primary Objective such that 4 mg and 2mg will be tested as co-primary objectives | Aligned the Primary Objective to support global regulatory feedback that require 2 mg and 4 mg to be tested on equal footing |
| 1. Synopsis | Added baricitinib 1-mg QD to the "Other Secondary Objective/Endpoint" evaluating the superiority of baricitinib compared to placebo, as measured by the proportion of patients achieving IGA of 0 or 1 with a ≥2-point improvement at Week 4 | Updated to align with all "Other<br>Secondary Objectives" |
| 2. Schedule of Activities | Removed wording about weighing tube with cap when dispensing rescue TCS | Decision made post-approval that the sponsor will take a baseline weight of full TCS tubes that are centrally supplied by the sponsor, instead of requiring the sites to weigh each full tube upon dispensing |
| 2. Schedule of Activities | Footnote "n" in the Schedule of Activities: corrected Visit 12 to Visit 7 (Week 12) | Corrected error |
| 4. Objectives and | Moved the 2-mg dose from Key Secondary | Aligns with changes in Section 1 |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| Endpoints | to Primary Objective | |
| 4. Objectives and Endpoints | Added baricitinib 1-mg QD to the "Other Secondary Objective/Endpoint" evaluating the superiority of baricitinib compared to placebo, as measured by the proportion of patients achieving IGA of 0 or 1 with a ≥2-point improvement at Week 4 | Aligns with changes in Section 1 |
| 6.1 Inclusion Criteria | #[6a] changed to read oral systemic corticosteroids | Clarified to distinguish between oral systemic corticosteroids versus parenteral corticosteroids administration which is covered in Exclusion Criterion #[17c] |
| 6.1. Inclusion Criteria | [7c]: deleted criterion "topical JAK inhibitor (e.g., tofacitinib or ruxolitinib) and/or any other investigative topical treatments" | This Inclusion Criterion was redundant since topic is already covered in Exclusion Criterion #[33], which has a broader time window. |
| 6.2. Exclusion Criteria | #[17b]: added wording "less than 4 weeks prior to randomization" for prior treatment with any oral JAK inhibitor | Since several oral JAK inhibitors are under development and discontinuation was most likely due to study participation completion and not adverse effects it was determined to allow prior use with a 4-week washout restriction. |
| 6.2. Exclusion Criteria | #[17e]: added criterion: "probenecid at the time of randomization (Visit 2) that cannot be discontinued for the duration of the study" | Co-administration of probenecid (an OAT3 inhibitor with strong inhibition potential) with baricitinib resulted in approximately a 2-fold increase in AUC(0-∞) with no change in tmax or Cmax of baricitinib. Thus, exclusion added to prohibit co-administration. |
| 6.2 Exclusion Criteria | #[20]: added "if participating in the trial at end of sentence | Added to clarify that the investigator is not evaluating the risk to the patient of the surgical procedure, rather the risk of participating in the trial. |
| 6.2 Exclusion Criteria | #[25a]: changed wording for cervical carcinoma in situ from "has been resected" to "has been appropriately treated" #[25b]: changed wording for basal cell or squamous epithelial skin cancers from "have been completely resected" to "have been appropriately treated" | Updated wording to address alternative treatment options available other than resection (e.g. surgical curettage and cautery, cryotherapy). |
| 6.2 Exclusion Criteria | #[31]: Removed "including use of data collection devices" | Revised in order to allow for some needed flexibility with the use of daily data collection devices (e.g. actigraphy) |
| 7.1.2. Medical Devices | Instructions for use on the wearing of actigraphy devices was revised and language was added to state that if not worn | Revised in order to allow for some needed flexibility with the use of |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| | as instructed that not considered a protocol violation | patients are allowed to remove the device if needed (e.g. showering); thus revised protocol language that previously stated "One will be worn on the wrist at all times" and added the statement that if not worn as instructed that it won't be considered a protocol violation. |
| 7.2. Method of Treatment<br>Assignment | Removed North America from region stratification | The US is no longer participating in this study and since they were the largest contributor to the NA region, this region was removed. |
| 7.7.1. Prohibited<br>Medications and<br>Procedures | Added 3 new subheader titles and reorganized and reordered existing bullets beneath each as appropriate | Done to clarify which prohibited medications would or would not require temporary interruption or permanent discontinuation of IP. |
| | Probenecid was added as a prohibited medication requiring temporary discontinuation of IP | Co-administration of probenecid (an OAT3 inhibitor with strong inhibition potential) with baricitinib resulted in approximately a 2-fold increase in AUC(0-\infty) with no change in tmax or Cmax of baricitinib. |
| 7.7.2. Permitted Medications and Procedures | Removed "prescription" with regards to use of emollients | Reimbursement for some non-additive emollients may require a prescription in some countries; thus to avoid these country specific differences, the term prescription was removed. |
| 7.7.3. Rescue Therapy | Section revised to incorporate language regarding additional options to supply equivalent potency TCS options (in addition to triamcinolone and hydrocortisone) | Due to potential supply issues, revisions were made to allow for other potential supply options for low-to-mid potency TCS options. |
| 7.7.3. Rescue Therapy | Added bullet point stating that topical therapy is not to be applied before study procedures | Application of topical therapies could impact adequate assessment of skin dryness thus clarification added in regards to application of topical rescue therapy on day of study visits. |
| 8.1.1. Temporary Interruption from Investigational Product | Table JAHL.4: last row wording modified to state "After evaluation and institution of appropriate treatment of VTEb." Removed "and resolution" | Criterion of "resolution of VTE" is not routinely assessed in clinical practice, thus language changed to a more objective measure. |
| 8.1.1. Temporary<br>Interruption from<br>Investigational Product | Table JAHL.4: related footnote b to VTE; revised the wording to align with changes listed above | Updated to match corresponding wording in table. |
| 8.1.1. Temporary Interruption from Investigational Product | Added text to refer reader to prohibited medications section (7.7.1) for details regarding temporary interruption of IP if a prohibited medication is taken | Added for clarification |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| 8.1.2. Permanent Discontinuation from Investigational Product | Deleted "or the patient's designee" | Removed since we are not allowing patients less than 18 year of age and we require patients to provide their own consent therefore not allowing consent from a patient's designee. |
| 8.1.2. Permanent Discontinuation from Investigational Product | Deleted "event" after VTE | Corrected error – use of "event" is redundant after VTE |
| 8.1.2. Permanent Discontinuation from Investigational Product | Added a final bullet to refer reader to prohibited medications section (7.7.1) for details regarding permanent discontinuation of IP if a prohibited medication is taken | Added for clarification |
| 8.2 Discontinuation from the Study | Deleted wording regarding a "patient's designee" | Removed since we are not allowing patients less than 18 year of age and we require patients to provide their own consent therefore not allowing consent from a patient's designee |
| 9.1.2.1. Eczema Area and<br>Severity Index Scores | Added reference | Updated based on feedback from a regulatory agency |
| 9.1.2.2. SCORing Atopic Dermatitis | Added references | Updated based on feedback from a regulatory agency |
| 9.5. Pharmacokinetics | Added wording that baseline laboratory samples are to be taken before administration of IP | Added for clarification |
| 10.1 Sample Size<br>Determination | Updated to reflect the change to co-primary objectives with no further implications on sample size. | Aligns with changes to the primary objective |
| 10.2 Populations for Analyses | Removed definition for safety follow-up population and added text to refer to SAP | The majority of patients are expected to enroll into extension study so safety follow-up population may not be useful for analysis. Further populations will be defined in the SAP. |
| 10.3.1 General Statistical<br>Considerations | Removed text that the Fisher exact test is only produced when logistic regression sample size requirements are not met | Both logistic regression and the Fisher exact test will be performed, regardless of logistic regression sample size requirements. |
| 10.3.1 General Statistical | Moved the 2-mg dose from Key Secondary | Aligns with changes to the primary |
| Considerations 10.3.4 Safety Analyses | Endpoint to Primary Endpoint Removed C-SSRS score from change from baseline analyses | Objective Correction of an error. C-SSRS will only be presented at the patient level as a listing. Further details will be in the SAP. |
| 11. References | References added to text updated in Reference list | Updated to align with Sections 9.1.2.1 and 9.1.2.2. |
| Appendix 1. Abbreviations and Definitions | Deleted US (United States) from list of abbreviations | Abbreviation not used in document |
| Appendix 1. Abbreviations | Added "deep vein thrombosis or pulmonary | Added for clarification |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| and Definitions | embolism" to definition of "VTE" | |
| Appendix 3. Study | Appendix 3.1.1 Informed Consent | Removed since we are not allowing |
| Governance Considerations | Removed "or legal representative" from second bullet point | patients less than 18 year of age and<br>we require patients to provide their<br>own consent therefore not allowing |
| | Removed text "A legal representative must give informed consent for a child to participate in this study" | consent from a legal representative. |

#### **Revised Protocol Sections**

Note: Deletions have been identified by strikethroughs.

Additions have been identified by the use of <u>underscore</u>.

#### Protocol cover page:

# Protocol I4V-MC-JAHL(a) A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Baricitinib in Adult Patients with Moderate to Severe Atopic Dermatitis

#### BREEZE-AD1

EudraCT Number: 2017-000870-12

#### 1. Synopsis

#### **Rationale:**

. . .

The pathogenesis of AD is thought to be modulated through thymic stromal lymphopoietin (TSLP), interleukin (IL)-13, <u>IL-4</u>, IL-5, IL-22, and IL-31, many of which activate receptors with downstream signaling through intracellular JAK1/JAK2/TYK2 (Nomura and Kabashima 2015)

. . .

| Objectives | Endpoints |
|---|---|
| Primary | |
| To test the hypothesis that baricitinib 4-mg QD or | <ul> <li>Proportion of patients achieving IGA of 0 or 1 with</li> </ul> |
| <u>baricitinib 2-mg QD</u> is superior to placebo in the | a ≥2-point improvement at Week 16. |
| treatment of patients with moderate to severe AD. | |
| Key Secondary | |
| These are prespecified objectives that will be adjusted j | for multiplicity |
| To test the hypothesis that baricitinib 2 mg QD or | <ul> <li>Proportion of patients achieving IGA of 0 or 1 with</li> </ul> |
| baricitinib 1-mg QD is superior to placebo in the | a ≥2-point improvement at Week 16. |
| treatment of patients with moderate to severe AD. | |

. . .

| Other Secondary Objectives | |
|---|---|
| These are prespecified objectives that will not be adjust | ted for multiplicity. |
| To test the hypothesis that baricitinib 1-mg QD, 2-mg | <ul> <li>Proportion of patients achieving IGA of 0 or 1 with</li> </ul> |
| QD, or 4-mg QD is superior to placebo in the | a ≥2-point improvement at Week 4. |
| treatment of patients with moderate to severe AD. | |

#### 2. Schedule of Activities

Table JAHL.1. I4V-MC-JAHL Schedule of Activities

| | Screening | Double-Blind, Placebo-Controlled | | | | Post-treatment<br>Follow-Up | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Period 1 | | | | Perio | d 2 | | | Period 3 |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 801a |
| Weeks from Randomization | | 0 | 1 | 2 | 4 | 8 | 12 | 16 or ET | |
| Days from Randomization | | 0 | 7 | 14 | 28 | 56 | 84 | 112 | |
| Visit tolerance interval (days) | -8 to -35 | | ±2 | ±2 | ±2 | ±4 | ±4 | ±4 | 28 ± 4 after last<br>dose |
| Procedure | | | | | | | | | |
| Dispense <del>and weigh (tube with eap)</del> rescue TCSh | | | X | X | X | X | X | X | |

...

| | Screening | Double-Blind, Placebo-Controlled | | | | | | Post-treatment<br>Follow-Up | |
|---|---|---|---|---|---|---|---|---|---|
| | Period 1 | Period 2 | | | | | Period 3 | | |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 801a |
| Weeks from Randomization | | 0 | 1 | 2 | 4 | 8 | 12 | 16 or ET | |
| Days from Randomization | | 0 | 7 | 14 | 28 | 56 | 84 | 112 | |
| Visit tolerance interval (days) | -8 to -35 | | ±2 | ±2 | ±2 | ±4 | ±4 | ±4 | 28 ± 4 after last<br>dose |
| Procedure | | | | | | | | | |
| Lipids (fasting) <sup>m</sup> | | X | | | | | X | Xn | X |

 $_{\rm n}$   $\,$  Only required for patients completing an ETV prior to completion of Visit  $\underline{127}$  (Week 12).

#### 4. Objectives and Endpoints

#### Table JAHL.2. Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| To test the hypothesis that baricitinib 4-mg QD or | <ul> <li>Proportion of patients achieving IGA of 0 or 1</li> </ul> |
| baricitinib 2-mg QD is superior to placebo in the | with a ≥2-point improvement at Week 16. |
| treatment of patients with moderate to severe AD. | |
| Key Secondary | |
| These are prespecified objectives that will be adjusted | for multiplicity |
| To test the hypothesis that baricitinib 2 mg QD or | Proportion of patients achieving IGA of 0 or 1 |
| baricitinib 1-mg QD is superior to placebo in the | with a ≥2-point improvement at Week 16. |
| treatment of patients with moderate to severe AD. | |

. . .

| Other Secondary Objectives | |
|---|---|
| These are prespecified objectives that will not be adjusted for multiplicity. | |
| To test the hypothesis that baricitinib 1-mg QD, | <ul> <li>Proportion of patients achieving IGA of 0 or 1</li> </ul> |
| 2-mg QD, or <del>baricitinib</del> 4-mg QD is superior to | with a ≥2-point improvement at Week 4 |
| placebo in the treatment of patients with moderate | |
| to severe AD. | |

#### 6.1. Inclusion Criteria

#### **Type of Patient and Disease Characteristics**

- [6] agree to discontinue use of the following excluded medications/treatments for at least 4 weeks prior to randomization (Visit 2) and throughout the study:
  - a. oral systemic corticosteroids and leukotriene inhibitors

. . .

[7] agree to discontinue use of the following excluded medications for at least 2 weeks prior to randomization (Visit 2) and throughout the study:

. . .

e Topical JAK inhibitor (e.g., tofacitinib or ruxolitinib) and/or any other investigative topical treatments.

#### 6.2. Exclusion Criteria

Patients will be excluded from study enrollment if they meet any of the following criteria:

#### **Medical Conditions Related to Atopic Dermatitis**

- [17] have been treated with the following therapies:...
  - b received prior treatment with any oral JAK inhibitor (e.g., tofacitinib, ruxolitinib) less than 4 weeks prior to randomization

e. probenecid at the time of randomization (Visit 2) that cannot be discontinued for the duration of the study

#### **Medical Conditions in General**

. . .

[20] have had any major surgery within 8 weeks prior to screening or will require major surgery during the study that, in the opinion of the investigator in consultation with Lilly or its designee, would pose an unacceptable risk to the patient if participating in the trial.

. .

- [25] have a history of lymphoproliferative disease; or have signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly; or have active primary or recurrent malignant disease; or have been in remission from clinically significant malignancy for less than 5 years.
  - a. Patients with cervical carcinoma in situ that has been <u>appropriately treated</u> resected with no evidence of recurrence or metastatic disease for at least 3 years may participate in the study.
  - b. Patients with basal cell or squamous epithelial skin cancers that have been appropriately treated completely resected with no evidence of recurrence for at least 3 years may participate in the study.

#### **Other Exclusions**

[31] are unable or unwilling to make themselves available for the duration of the study and/or are unwilling to follow study restrictions/procedures, including use of data collection devices.

#### 7.1.2. Medical Devices

An actigraphy device, a hypoallergenic device worn on the wrist, will be used to collect sleep/wake patterns and quantify nocturnal scratching events. Each patient will be dispensed 2 actigraphy devices. One <u>shouldwill</u> be worn on the wrist <u>during waking hoursat all times</u> and the other <u>shouldwill</u> be worn only during hours of sleep. Patients will be provided instructions on use and when to bring the devices back to study site based on Schedule of Activities (Section 2). If devices are not worn as instructed, it will not be considered a protocol violation.

#### 7.2. Method of Treatment Assignment

Patients who meet all criteria for enrollment will be randomized in a 2:1:1:1 ratio (placebo, baricitinib 1 mg; baricitinib 2 mg; baricitinib 4 mg) to double blind treatment at Visit 2 (Week 0). Randomization will be stratified by geographic region (North America [NA], Europe [EU], Japan [JPN], rest of world [ROW]) and disease severity at baseline (IGA 3 vs. 4).

#### 7.7.1. Prohibited Medications and Procedures

#### <u>Prohibited Medications and Procedures Not Requiring Interruption of Investigational</u> Product

The following therapies will not be <u>allowed</u>permitted during the course of the study <u>and</u>, <u>if taken</u> by or administered to the patient, the prohibited therapy must be discontinued.

- TCS, TCNIs (e.g., tacrolimus and pimecrolimus), or topical PDE 4 inhibitor (i.e., crisaborole) except when given as rescue therapy as described in Section 7.7.3.
- topical antihistamines or sedating, systemic antihistamines including, but not limited to, alimemazine, chlorphenamine, clemastine, cyproheptadine, diphenhydramine, hydroxyzine, ketotifen, and promethazine
- leukotriene inhibitors (e.g., montelukast [Singulair], zafirlukast [Accolate], and zileuton [Zyflo])
- allergen immunotherapy
- phototherapy including PUVA (psoralen and ultraviolet A), ultraviolet B, tanning booth and excimer laser
- bleach baths

#### **Prohibited Medications Requiring Temporary Interruption of Investigational Product**

The following therapies will not be allowed during the course of the study and, if taken by or administered to the patient, temporary interruption of investigational product is required.

- live vaccines (including Bacillus Calmette-Guérin [BCG] or herpes zoster), (see Exclusion Criterion [27])
  - o For BCG vaccination, investigational product should be temporarily interrupted for 12 weeks.
  - o <u>For herpes zoster vaccination</u>, investigational product should be temporarily interrupted for 4 weeks.
- probenecid: if a patient is inadvertently started on probenecid, IP should be temporarily interrupted, and can be resumed after patient has discontinued probenecid. If a patient is not able to discontinue probenecid, then IP should be permanently discontinued

#### Prohibited Medications Requiring Permanent Discontinuation of Investigational Product

- systemic corticosteroids
- any systemic therapy, investigational or commercial (approved or off label use), used for the treatment of AD or symptoms of AD (except for antihistamines, as specified above)
- other JAK inhibitors (e.g., tofacitinib and ruxolitinib)

 systemic immunosuppressive/immunomodulatory substances, including, but not limited to, cyclosporine, methotrexate, mycophenolate mofetil, interferon γ, azathioprine, or biologic agents

Note: In the event that these prohibited medications were inadvertently used, agreement and documentation to continue investigational product must be sought from sponsor.

#### 7.7.2. Permitted Medications and Procedures

Treatment with concomitant AD therapies during the study is permitted only as described below.

• Daily use of emollients is required as background treatment. Prescription moisturizers or mMoisturizers with additives such as antiprurities or antiseptics are not permitted. If daily applications are missed, it will not be considered a protocol violation.

#### 7.7.3. Rescue Therapy

. .

#### Choice of rescue therapy treatment

- Triamcinolone 0.1% cream and/or hydrocortisone 2.5% ointment. Where possible, Bboth of these treatments will be eentrally supplied by the sponsor. In the event countries where providing 1 or both of these topical formulations is not possible, an alternate, equivalent potency TCS cream and/or ointment that is in line with local practices can be considered; however, it will not may be provided centrally by the sponsor. TCS use, supplied by the sponsor, should be recorded via weight of returned tubes as indicated in the Schedule of Activities (Section 2).
  - o In the event that the sponsor is unable to supply TCS, commercially available triamcinolone 0.1% cream and/or hydrocortisone 2.5% ointment may be supplied by the sites. Where providing triamcinolone 0.1% cream and/or hydrocortisone 2.5% ointment is not possible, an equivalent-potency TCS cream and/or ointment that is in line with local practices can be supplied. Refer to Appendix 7 for guidance on potency equivalence.
  - O If the TSC supplied by the sponsor is not considered suitable for an individual patient, an equivalent-potency TCS cream and/or ointment that is in line with local practices can be supplied by the sites. Refer to Appendix 7 for guidance on potency equivalence.
- Investigators may also select to use TCNIs and/or crisaborole where approved, although use of either during the study is neither encouraged nor provided. If TCNIs are prescribed, use should be limited to problem areas only (e.g., face, neck, skin folds, genital areas, etc.).
- On the days of study visits, topical therapy should not be applied before the patient has undergone all study procedures and clinical evaluations in order to allow adequate assessment of skin dryness

#### 8.1.1. Temporary Interruption from Investigational Product

#### Table JAHL.4. Criteria for Temporary Interruption of Investigational Product

| Hold Investigational Product if the Following Laboratory Test Results or Clinical Events Occur: | Investigational Product May Be Resumed When: |
|---|---|
| WBC count <2000 cells/μL | WBC count ≥2500 cells/μL |
| $(<2.00x10^3/\mu L \text{ or } <2.00 \text{ GI/L})$ | $(\ge 2.50 \times 10^3 / \mu L \text{ or } \ge 2.50 \text{ GI/L})$ |
| Clinical features of VTE (such as deep vein thrombosis or | After evaluation and institution of appropriate |
| pulmonary embolism) are presenta | treatment and resolution of VTEb |

Abbreviations: ALT = alanine aminotransferase; ANC = absolute neutrophil count; AST = aspartate aminotransferase; eGFR = estimated glomerular filtration rate; IP = investigational product; ULN = upper limit of normal; VTE = venous thromboembolic event; WBC = white blood cell.

- <sup>a</sup> Evaluate promptly and institute appropriate treatment. If upon evaluation VTE is ruled out and no other temporary or permanent discontinuation criteria are met, then IP may be resumed.
- b If upon after evaluation and institution of treatment resolution the investigator deems that the patient is still at significant risk, or if this would constitute a second VTE for the patient, then IP should be discontinued permanently

Although temporary interruption of investigational product is not a requirement at times of increased potential risk of VTE (e.g., surgery, significant air travel, or other situations involving prolonged immobilization) we recommend following appropriate VTE prophylaxis guidelines to help manage the VTE risk under these circumstances.

For specific guidance on temporary interruption of IP after use of a prohibited medication, please refer to Section 7.7.1 (Prohibited Medications and Procedures).

#### 8.1.2. Permanent Discontinuation from Investigational Product

Investigational product should be permanently discontinued if the patient or the patient's designee requests to discontinue investigational product.

. . .

In addition, patients will be discontinued from investigational product in the following circumstances:

- pregnancy
- malignancy (except for successfully treated basal or squamous cell skin carcinoma)
- hepatitis B virus DNA is detected with a value above limit of quantitation or 2 sequential tests return a value of below the limit of quantitation (see Section 9.4.8).
- develop a second VTE event
- <u>certain prohibited medications are taken per Section 7.7.1 (Prohibited Medications and Procedures).</u>

#### 8.2. Discontinuation from the Study

. . .

Some possible reasons that may lead to permanent discontinuation include the following:

- ...
- patient decision
  - o The patient or the patient's designee, for example, parents or legal guardian, requests to be withdrawn from the study.

#### 9.1.2.1. Eczema Area and Severity Index Scores

The EASI assesses extent of disease at 4 body regions and measures 4 clinical signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3. The EASI confers a maximum score of 72. The EASI evaluates 2 dimensions of AD: disease extent and clinical signs (Hanifin et al. 2001).

#### 9.1.2.2. SCORing Atopic Dermatitis

The SCORing Atopic Dermatitis (SCORAD) index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness. The SCORAD index also assesses subjective symptoms of pruritus and sleep loss. These 3 aspects: extent of disease, disease severity, and subjective symptoms combine to give a maximum possible score of 103 (Stalder et al. 1993; Kunz et al. 1997; Schram et al. 2012).

#### 9.5. Pharmacokinetics

A venous blood sample will be drawn at the times indicated in the Schedule of Activities (Section 2) (Weeks 0 [first dose, 2 samples], 4, 8, 12, and 16). These blood samples will be used to determine the plasma concentrations of baricitinib using a validated liquid chromatography tandem mass spectrometry method. Blood samples that will be used for other laboratory assessments (chemistry, hematology, etc.) should be drawn at approximately the same time as the samples drawn to determine plasma concentrations of baricitinib. The timing will be as follows:

• At Visit 2 (Week 0), <u>baseline laboratory samples should be taken before</u> <u>administration of investigational product.</u> <u>pPatients will take their investigational product in the clinic, and PK samples will be drawn 15 minutes and 1 hour postdose.</u>

#### 10.1. Sample Size Determination

Study JAHL will aim to enroll approximately 600 patients ≥18 years of age. The proposed sample size will ensure a >90% power to detect an absolute difference of 20% between the baricitinib 4-mg and placebo treatment groups and the baricitinib 2-mg and placebo treatment groups, each using a 2-sided alpha of 0.025, assuming a 10% placebo response rate for the primary endpoint using a 2 sided alpha of 0.05.

#### 10.2. Populations for Analyses

. . .

Safety analyses for the post treatment Follow up Period will be conducted on the follow up population, defined as all randomized patients who received at least 1 dose of investigational product and have entered the post treatment Follow Up Period.—Further details of other populations will be described in the SAP. Patients will be analyzed according to the dosing regimen to which they were assigned in the Treatment Period.

#### 10.3.1. General Statistical Considerations

•••

All tests of treatment effects will be conducted at a 2 sided alpha level of 0.05, unless otherwise stated. Treatment comparisons of discrete efficacy variables between baricitinib and placebo will be made using a logistic regression analysis with region, disease severity, and treatment group in the model. The percentages, difference in percentages, and 95% confidence interval (CI) of the difference in percentages will be reported. Treatment by region interaction will be added to the logistic regression model of the primary and key secondary variables as a sensitivity analysis. If this interaction is significant at a 2 sided 0.1 level, further inspection will be used to assess whether the interaction is quantitative (i.e., the treatment effect is consistent in direction but not size of effect) or qualitative (the treatment is beneficial for some but not all regions). When logistic regression sample size requirements are not met (<5 responders in any category for any factor), tThe p-value from the Fisher exact test will also be produced instead of the odds ratio and CI.

...

#### **Adjustment for Multiple Comparisons:**

. .

The following is a list of primary and key secondary endpoints to be tested:

#### Primary:

- proportion of baricitinib 4-mg patients achieving IGA of 0 or 1 and ≥2-point improvement from baseline at Week 16.
- proportion of baricitinib 2-mg patients achieving IGA of 0 or 1 and ≥2-point improvement from baseline at Week 16.

#### Key Secondaries:

• proportion of baricitinib-2 mg or 1-mg patients achieving IGA of 0 or 1 with a ≥2-point improvement at Week 16.

#### 10.3.4. Safety Analyses

٠..

Observed values and changes from baseline (predose or screening if missing) for vital signs and physical characteristics will be descriptively summarized by treatment group and time point. Change from baseline to postbaseline in vital signs, C SSRS score, and body weight will be analyzed using ANCOVA with treatment and baseline value in the model.

#### 11. References

. . .

Hanifin JM, Thurston M, Omoto M, Cherill R, Tofte SJ, Graeber M. The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. EASI Evaluator Group. *Exp Dermatol*. 2001;10(1):11-18.

. . .

Kunz B, Oranje A, Labrèze L, Stadler JF, Ring J, Taïeb A, Clinical Validation and Guidelines for the SCORAD Index: Consensus Report of the European Task Force on Atopic Dermatitis. <u>Dermatology</u>. 1997;195(1):10-19.

. . .

Schram ME, Spuls PI, Leeflang MM, Lindeboom R, Bos J, Schmitt J. EASI, (objective) SCORAD and POEM for atopic eczema:responsiveness and minimal clinically important difference. *Allergy*. 2012;67:99-106.

. . .

Stalder JF, Taieb A, Atherton DJ, et al. for the European Task Force on Atopic Dermatis.

Severity scoring of atopic dermatitis: the SCORAD index. Consensus Report of the European Task Force on Atopic Dermatitis. *Dermatology*. 1993;186(1):23-31.

#### Appendix 1. Abbreviations and Definitions

| Term | Definition |
|---|---|
| US | United States |
| VTE | venous thromboembolic event (deep vein thrombosis or pulmonary embolism) |

#### Appendix 3.1.1. Informed Consent

The investigator is responsible for ensuring the following:

- that the patient understands the potential risks and benefits of participating in the study.
- that informed consent is given by each patient or legal representative. This includes obtaining the appropriate signatures and dates on the informed consent form (ICF) prior to the performance of any protocol procedures and prior to the administration of investigational product.
- answering any questions the patient may have throughout the study and sharing in a timely manner any new information that may be relevant to the patient's willingness to continue his or her participation in the trial.

A legal representative must give informed consent for a child to participate in this study. In addition to informed consent given by the legal representative, the child may be required to give documented assent, if capable.

Leo Document ID = d33530cb-1960-4b47-8354-2212ad3648f7

Approver: PPD

Approval Date & Time: 15-Dec-2017 15:05:07 GMT

Signature meaning: Approved

Approver: PPD

Approval Date & Time: 15-Dec-2017 18:16:50 GMT

Signature meaning: Approved